CLINICAL TRIAL: NCT02592434
Title: EFFICACY, SAFETY AND TOLERABILITY OF TOFACITINIB FOR TREATMENT OF POLYARTICULAR COURSE JUVENILE IDIOPATHIC ARTHRITIS (JIA) IN CHILDREN AND ADOLESCENT SUBJECTS
Brief Title: Efficacy Study Of Tofacitinib In Pediatric JIA Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921104; 2015-001438-46 (EudraCT Number); PROPEL STUDY (Other: Alias Study Number); PROPEL (Other: Alias Study Number)
Record Dates: First submitted 2015-08-14; First posted 2015-10-30 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Arthritis; Pediatric; Long-term; JIA; polyarticular; CP-690,550; tofacitinib; Xeljanz
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — tofacitinib; S-Adenosylmethionine; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CP-690,550 (Experimental): Treatment arm: Tofacitinib tablets or solution, according to subjects' body weights
  Interventions: Drug: CP-690,550 (tofacitinib)
- Placebo (Placebo Comparator): Control arm: matching placebo tablets or solution for tofacitinib
  Interventions: Other: placebo

INTERVENTIONS:
Drug: CP-690,550 (tofacitinib) — During the open label run in phase, all subjects will receive active tofacitinib oral tablets or oral solution twice daily (BID) orally, at a dosage based on the subject's body weight as specified below.
  During the double blind, placebo controlled phase, subjects will receive either active tofacitinib oral tablets/oral solution or matching placebo oral tablets/oral solution, twice daily (BID), at a dosage specified below.
  Body Weight (Dosage in tablet [BID] or solution [BID]):
  5<7kg (2mg or 2mL); 7<10kg(2.5mg or 2. mL); 10 <15kg (3mg or 3mL); 15<25kg (3.5mg or 3.5mL); 25<40kg (4mg or 4mL); 40kg (5 mg or 5 ml).
  Oral solution (1 mg/mL) is used for subjects <40 kg. Oral tablets (5 mg) are used for subjects >=40 kg.
  Other Names: Matching placebo to tofacitinib (same tablet or solution as the active arm).
  Arms: CP-690,550
Other: placebo — matching placebo tablet or solution for tofacitinib
  Other Names: Placebo for tofacitinib
  Arms: Placebo

SUMMARY:
Evaluate efficacy, safety and tolerability of tofacitinib in pediatric JIA patients.

DETAILED DESCRIPTION:
This is a randomized withdrawal, double blind, placebo controlled study of pediatric subjects (2 to <18 years of age) with JIA. The primary objective is to compare the efficacy of tofacitinib versus placebo for the treatment of signs and symptoms of JIA at Week 26 of the double blind phase as measured by the percentage of subjects with disease flare (according to PRCSG/PRINTO Disease Flare criteria) after Week 18 of the open label run in phase.All eligible subjects enrolled in the study will initially receive open label tofacitinib for 18 weeks (run in phase). At the end of the 18 week run in phase, only subjects who achieve at least a JIA ACR 30 response will be randomized to the 26 week double blind, placebo controlled phase. Subjects who do not achieve a JIA ACR 30 response at this time point will be discontinued from the study. In addition, subjects who experience a single episode of disease flare at any time during the study (including the open label run in and double blind phase) will also be discontinued from the study. All subjects participating in this study, including those discontinued from the study, will have the option, if eligible (based on inclusion and exclusion criteria), of enrolling in the tofacitinib JIA long term extension study (A3921145).

Subjects who are eligible for the 26 week double blind phase will be randomized (1:1 ratio) to either active tofacitinib or placebo. For subjects with polyarticular course JIA (ie, extended oligoarthritis, polyarthritis RF+, polyarthritis RF , systemic JIA with active arthritis but without active systemic features), randomization will be stratified by JIA category and baseline CRP (normal, above normal). For subjects with psoriatic and enthesitis related arthritis, randomization will be stratified by JIA category.

Approximately 210 subjects will be enrolled in the open label run in phase. Among subjects with polyarticular course JIA, stratification will target at least 50% with a baseline CRP above the upper limit of normal. The first cohort (ie, polyarticular course JIA) will have at least 170 subjects enrolled in the run in phase with the minimum number of JIA categories as follows: 24 with extended oligoarthritis, 20 with polyarthritis RF+, 62 with polyarthritis RF-, and no minimum for subjects with systemic JIA with active arthritis but without active systemic features. Additional cohorts (ie, psoriatic and enthesitis related arthritis) will include a minimum of 20 subjects with psoriatic arthritis, and 20 subjects with enthesitis related arthritis. The overall target minimum number of subjects to be enrolled in the study by age is as follows: 20 subjects 2 to <6 years, 20 subjects 6 to <12 years, and 20 subjects 12 to <18 years. The duration of subject participation among those who complete the study (without discontinuation) is expected to be approximately 44 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 2 to <18 years.
2. Must meet International League Against Rheumatism (ILAR) JIA diagnostic criteria for one of the following categories with active disease for at least 6 weeks:

   * Extended oligoarthritis;
   * Polyarthritis (RF+);
   * Polyarthritis (RF-);
   * Systemic JIA with active arthritis but without active systemic features in the prior 6 months and at the time of enrollment;
   * Psoriatic arthritis;
   * Enthesitis related arthritis. Subjects with polyarticular course JIA (ie, extended oligoarthritis, polyarthritis RF+, polyarthritis RF , systemic JIA with active arthritis but without active systemic features) must have a minimum of 5 active joints (an active joint is defined as a joint with swelling or, in the absence of swelling, limited range of motion accompanied by either pain on motion or tenderness) at screening and baseline to be eligible for study entry.

   Subjects with psoriatic or enthesitis related arthritis must have a minimum of 3 active joints (an active joint is defined as a joint with swelling or, in the absence of swelling, limited range of motion accompanied by either pain on motion or tenderness) at screening and baseline to be eligible for study entry.

   Treatment with stable doses of a Non Steroidal Anti inflammatory Drug (NSAID) and/or a stable dose of an oral glucocorticoid, and/or a stable dose of methotrexate is permitted.

   For subjects receiving an oral glucocorticoid: Glucocorticoids may be administered at a maximum dose of 0.2 mg of prednisone equivalent per kilogram per day or 10 mg per day for ≥ 2 weeks before baseline, whichever is lower.

   For subjects receiving methotrexate (MTX) treatment: MTX may be administered either orally or parenterally at doses not to exceed 25 mg/wk or 20 mg/m2/week (whichever is lower); participants must have taken MTX for 3 months and be at a stable dose for at least 6 weeks before baseline. Subjects taking MTX must be taking folic acid or folinic acid in accordance with local standards.

   For subjects with psoriatic arthritis, the following topical treatments for psoriasis are allowed: non medicated emollients for use over the whole body; topical steroids including hydrocortisone and hydrocortisone acetate ≤1% for the palms, soles, face, and intertriginous areas only; tar, salicylic acid preparations, and shampoos free of corticosteroids are permitted only for the scalp
3. Inadequate response or intolerance to at least one Disease Modifying Anti Rheumatic Drug (DMARD), which may include MTX or biologic agents; in the case of ERA and psoriatic arthritis, inadequate response to Non Steroidal Anti Inflammatory Drugs (NSAIDs).
4. No evidence or history of untreated or inadequately treated active or latent tuberculosis (TB) infection as evidenced by the following:

   1. A negative QuantiFERON ®TB Gold In Tube test performed within the 3 months prior to screening. A negative purified protein derivative (PPD) test can be substituted for the QuantiFERON® TB Gold In Tube test only if the central laboratory is unable to perform the test or cannot determine the results to be positive or negative and the Pfizer medical monitor is informed and agrees on a case by case basis.
   2. Chest radiograph without changes suggestive of active tuberculosis (TB) infection within 3 months prior to screening is recommended and should be performed according to local standards of care or country-specific guidelines.
   3. No history of either untreated or inadequately treated latent or active TB infection.

   If a subject has previously received an adequate course of therapy for either latent (9 months of isoniazid in a locale where rates of primary multi drug resistant TB infection are <5% or an acceptable alternative regimen) or active (acceptable multi drug regimen) TB infection, neither a PPD test nor a QuantiFERON-Gold®TM test need be obtained. A chest radiograph should be obtained if not done within the 3 months prior to screening. To be considered eligible for the study, the chest radiograph must be negative for active tuberculosis infection.

   A subject who is currently being treated for latent TB infection can only be enrolled with confirmation of current incidence rates of multi-drug resistant TB infection, documentation of an adequate treatment regimen, and prior approval of the Sponsor.
5. Fertile males and females who are, in the opinion of the investigator, sexually active and at risk for pregnancy with their partner(s) must be willing and able to use a highly effective method of contraception as outlined in this protocol during the study and for at least 28 days after the last dose of study medication.

6 Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

7. Evidence of a personally signed and dated Informed Consent document and Assent document (as appropriate) indicating that the subject and a legally acceptable representative/parent(s)/legal guardian has been informed of all pertinent aspects of the study.

Exclusion Criteria

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Previous JIA treatment with tofacitinib.
2. Systemic JIA (sJIA) with active systemic features (including subjects with characteristic sJIA fever and rash or serositis within 6 months of enrollment).
3. Persistent oligoarthritis.
4. Undifferentiated JIA.
5. Infections:

   1. Chronic infections;
   2. Any infection requiring hospitalization, parenteral antimicrobial therapy or judged to be opportunistic by the investigator within the 6 months prior to the first dose of study drug;
   3. Any treated infections within 2 weeks of Baseline visit;
   4. A subject know to be infected with Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C;
   5. History of infected joint prosthesis with prosthesis still in situ.
6. History of recurrent (more than one episode) herpes zoster or disseminated (at least one episode) herpes zoster, or disseminated (at least one episode) herpes simplex.
7. Active uveitis (according to SUN criteria) within 3 months of enrollment.
8. Blood dyscrasias, including:

   1. Hemoglobin <10 g/dL or Hematocrit <33%;
   2. White Blood Cell count <3.0 x 109/L;
   3. Neutrophil count <1.2 x 109/L;
   4. Platelet count <100 x 109/L;
   5. Lymphocyte count <0.75 x 109/L.
9. Estimated glomerular filtration rate [GFR] <40 mL/min/1.73 m2 at Screening. GFR will be calculated by the central lab using the bedside Schwartz formula.
10. Current or recent history of uncontrolled clinically significant renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurologic disease.
11. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥1.5 times the upper limit of normal.
12. History of any other rheumatologic disease, other than Sjogren's syndrome..
13. History or current symptoms suggestive of lymphoproliferative disorders (eg, Epstein Barr Virus [EBV] related lymphoproliferative disorder, lymphoma, leukemia, or signs and symptoms of current lymphatic disease).
14. Vaccinated or exposed to a live or attenuated vaccine within the 6 weeks prior to the first dose of study drug, or is expected to be vaccinated or to have household exposure to these vaccines during treatment or during the 6 weeks following discontinuation of study drug.
15. Subjects without documented evidence of having received at least one dose of the varicella vaccine in countries where the vaccine is approved and standard of care or those who do not have evidence of prior exposure to varicella zoster virus (VZV) based on serological testing (ie, VZV IgG Ab).
16. Current malignancy or history of any malignancy with the exception of adequate treated or excised basal cell or squamous cell or cervical cancer in situ.
17. Subjects who have previously failed more than 3 biologic therapies (with different mechanisms of action) for JIA.
18. Subjects with a first degree relative with a hereditary immunodeficiency; IgA deficiency not exclusionary.
19. Recent (within 28 days prior to first dose of study drug) significant trauma or major surgery.
20. Subjects receiving potent and moderate CYP3A4 inhibitors or inducers.
21. Prior treatment with non B cell specific lymphocyte depleting agents/therapies (eg, almetuzumab [CAMPATH], alkylating agents [eg, cyclophosphamide or chlorambucil], total lymphoid irradiation, etc.). Subjects who have received rituximab or other selective B lymphocyte depleting agents (including experimental agents) are eligible if they have not received such therapy for at least 1 year prior to study baseline and have normal CD 19/20+ counts by FACS analysis.
22. Use of prohibited prescription or non prescription drugs and dietary supplements listed in Appendix 1 and Appendix 4 within the specified time frame prior to the first dose of study medication.
23. Herbal supplements must be discontinued at least 28 days prior to the first dose of study medication.
24. Use of certain biologic and non biologic DMARDs are disallowed at any time during this study (Appendix 1).
25. For subjects with PsA, oral and topical medications and alternative treatments that could affect psoriasis are prohibited (see Inclusion Criterion 2 for exceptions). This includes topical corticosteroids, tars, keratolytics, anthralin, vitamin D analogs, and retinoids which must be discontinued at least 2 weeks prior to first dose of study drug. Also prohibited is ultraviolet B (UVB) (narrowband or broadband) phototherapy that must be discontinued at least 2 weeks prior to first dose of study drug. Psoralens + ultraviolet A (UVA) phototherapy (PUVA) must be discontinued at least 4 weeks prior to first dose of study drug.
26. Subjects who are children of or related to investigational site staff members, site staff members otherwise supervised by the investigator, or Pfizer employees directly involved in the conduct of the study.
27. Participation in other studies involving investigational drug(s) within 4 weeks or 5 half lives (whichever is longer) prior to study entry and/or during study participation. Exposure to investigational biologics should be discussed with the Sponsor.
28. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
29. Pregnant or nursing females are excluded.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (101):
- United States (55):
  - Arkansas Children's Hospital - Attention: Jill Hernandez, Little Rock, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Loma Linda University Clinical Trial Center, Loma Linda, California
  - Loma Linda University Eye Institute, Loma Linda, California
  - Loma Linda University General Pediatric Clinic - Meridian, Loma Linda, California
  - Pediatric Specialty Team Centers of LLU Children's Hospital, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Pediatric Specialty Team Centers of LU Children's Hospital, San Bernardino, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Rady Children's Hospital Center for Pediatric Clinical Research, San Diego, California
  - Rady Children's Hospital Education and Office Building, San Diego, California
  - Rady Children's Hospital Research Pharmacy, San Diego, California
  - Rady Children's Hospital Rheumatology Clinic, San Diego, California
  - Connecticut Children's Medical Center -Pharmacy, Hartford, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - IDS Pharmacy Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta-Pediatric Research Center, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Specialty Services, Atlanta, Georgia
  - Augusta University Health Pharmacy, Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - IU Health Investigational Drug Services, Indianapolis, Indiana
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Tufts Medical Center Floating Hospital for Children, Boston, Massachusetts
  - Journey Clinic: Center for Children with Cancer and Blood Diseases, Uni. of Minnesota Medical Centre, Minneapolis, Minnesota
  - Pediatric Specialty Care Explorer Clinic, University of Minnesota, Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview IDS Pharmacy, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cohen Children's Medical Center of NY, Lake Success, New York
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Pharmacy Department, The Bronx, New York
  - Children's Specialty Center, Charlotte, North Carolina
  - Carolinas HealthCare System IDS Pharmacy, Charlotte, North Carolina
  - Pediatric Research, Charlotte, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Legacy Emanuel Medical Center - Inpatient Pharmacy, Portland, Oregon
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Specially for Children, Dell Children's Medical Center of Central Texas, Austin, Texas
  - Texas Children's Hospital - Clinical Care center, Houston, Texas
  - Texas Children's Hospital - Clinical Research Center, Houston, Texas
  - Texas Children's Hospital - Investigational Pharmacy, Houston, Texas
  - Texas Children's Hospital - Main Hospital, Houston, Texas
  - Texas Children's Hospital/Baylor College of Medicine - Feigin Center, Houston, Texas
  - PCH Pharmacy - Primary Children's Hospital - Pharmacy, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Argentina (3):
  - Instituto CAICI SRL, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Hospital Britanico de Buenos Aires, CABA
- Australia (2):
  - The Sydney Children's Hospital Network Westmead, Westmead, New South Wales
  - The Royal Children's Hospital, Parkville, Victoria
- UZ Leuven-Gasthuisberg, Leuven, Belgium
- Brazil (9):
  - SER - Servicos Especializados em Reumatologia, Salvador, Estado de Bahia
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - CMIP -Centro Mineiro de Pesquisa Ltda / Reumatocenter, Juiz de Fora, Minas Gerais
  - Hospital Pequeno Principe / A ssociacao Hospitalar de Protecao a Infancia, Curitiba, Paraná
  - Instituto de Pesquisa Pele Pequeno Principe, Curitiba, Paraná
  - Instituto de Puericultura e Pediatria Martagao Gesteira, Rio de Janeiro, Rio de Janeiro
  - Faculdade de Medicina da UNESP, Botucatu, São Paulo
  - SPDM- Associacao Paulista para o Desenvolvimento da Medicina-Hospital Sao Paulo, São Paulo
  - Instituto da Crianca do Hospital das Clinicas da FMUSP, São Paulo
- Canada (6):
  - Alberta Children's Hospital - Inpatient Pharmacy, Calgary, Alberta
  - Alberta Children's Hospital/University of Calgary, Calgary, Alberta
  - Children's & Women's Health Centre of B.C., Vancouver, British Columbia
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - McGill University Health Canter, Glen site, Pharmacy, Montreal, Quebec
  - McGill University Health Center, Glen Site, Center for Innovative Medicine, Montreal, Quebec
- Israel (3):
  - Rambam Health Care, Haifa
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba M.C Tel hashomer, Ramat Gan
- Mexico (5):
  - Clinica de Investigacion en Reumatologia y Obesidad, S.C., Guadalajara, Jalisco
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi S.C., San Luis Potosí City
  - Sociedad de Beneficencia Espanola, A.C., San Luis Potosí City
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
  - Unidad de Investigaciones Reumatologicas A.C., San Luis Potosí City
- Wojewodzki Szpital Dzieciecy im. J. Brudzinskiego, Bydgoszcz, Poland
- Russia (5):
  - FSAEI HE I.M. Sechenov First MSMU of Minzdrav of Russia (Sechenovskiy University), Moscow
  - FSAEI HE I.M Sechenov First MSMU of Minzdrav of Russia (Sechenovskiy University), Moscow
  - FSAI "NSPCCH" of Minzdrav of Russia, Moscow
  - FSBEI HE "St. Petersburg State Pediatric Medical University", Saint Petersburg
  - State Budgetary Healthcare Institution of Samara Region "Tolyatti City Clinical Hospital #5", Tolyatti
- Spain (2):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul Medeniyet University Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Umraniye Training and Research Hospital, Istanbul
  - Erciyes University Medical Faculty, Kayseri
- Ukraine (2):
  - Ivano-Frankivsk Regional Children's Clinical Hospital, Ivano-Frankivsk
  - Vinnytsia Regional Children's Clinical Hospital, Vinnytsia
- United Kingdom (2):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Birmingham Woman's and Children's NHS Foundation Trust, Birmingham, WEST Midlands

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Consolaro A, Ruperto N, Lovell DJ, Synoverska O, Abud-Mendoza C, Spindler A, Vyzhga Y, Alexeeva E, Chaitow J, Chiraseveenuprapund P, Lazariciu I, Stockert L, Cadatal MJ, Diehl A, Brunner HI; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Clinically Inactive Disease and Remission in Patients With Juvenile Idiopathic Arthritis Receiving Tofacitinib: Post Hoc Analysis of a Phase III Trial. J Rheumatol. 2025 Sep 1;52(9):919-926. doi: 10.3899/jrheum.2024-0536. PMID 40312101
- [Derived] Chang C, Vong C, Wang X, Hazra A, Diehl A, Nicholas T, Mukherjee A. Tofacitinib pharmacokinetics in children and adolescents with juvenile idiopathic arthritis. CPT Pharmacometrics Syst Pharmacol. 2024 Apr;13(4):599-611. doi: 10.1002/psp4.13104. Epub 2024 Jan 31. PMID 38298058
- [Derived] Ruperto N, Brunner HI, Synoverska O, Ting TV, Mendoza CA, Spindler A, Vyzhga Y, Marzan K, Grebenkina L, Tirosh I, Imundo L, Jerath R, Kingsbury DJ, Sozeri B, Vora SS, Prahalad S, Zholobova E, Butbul Aviel Y, Chasnyk V, Lerman M, Nanda K, Schmeling H, Tory H, Uziel Y, Viola DO, Posner HB, Kanik KS, Wouters A, Chang C, Zhang R, Lazariciu I, Hsu MA, Suehiro RM, Martini A, Lovell DJ; Paediatric Rheumatology International Trials Organisation (PRINTO) and Pediatric Rheumatology Collaborative Study Group (PRCSG). Tofacitinib in juvenile idiopathic arthritis: a double-blind, placebo-controlled, withdrawal phase 3 randomised trial. Lancet. 2021 Nov 27;398(10315):1984-1996. doi: 10.1016/S0140-6736(21)01255-1. Epub 2021 Nov 9. PMID 34767764
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921104

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib: Open-Label Phase: Participants received tofacitinib 5 mg tablets (for participants >= 40 kg body weight) or tofacitinib 5 mL oral solution (for participants <40 kg body weight), BID, orally for 18 weeks in open-label phase.
- Tofacitinib: Double Blind Phase: Participants who completed open-label phase and achieved at least a Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 response in open label phase, were randomized at Week 18 to receive tofacitinib tablets (for participants >=40 body weight) or oral solution (for participants <40 kg body weight), BID, in double-blind phase for additional 26 weeks (up to Week 44).
- Placebo: Participants who completed open-label phase and achieved at least a JIA ACR 30 response in open label phase, were randomized at Week 18 to receive placebo either as oral tablets, (for subjects >=40 body weight) or oral solution (for subjects <40 kg body weight), BID, in double-blind phase for additional 26 weeks (up to Week 44).
Period: Open-Label Phase (18 Weeks)
Arm/Group | Tofacitinib: Open-Label Phase | Tofacitinib: Double Blind Phase | Placebo
Started | 225 | 0 | 0
Treated | 225 | 0 | 0
Completed | 185 | 0 | 0
Not Completed | 40 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0
Not completed — Insufficient Clinical Response | 21 | 0 | 0
Not completed — Other | 3 | 0 | 0
Not completed — Protocol Deviation | 4 | 0 | 0
Period: Double Blind Phase (26 Weeks)
Arm/Group | Tofacitinib: Open-Label Phase | Tofacitinib: Double Blind Phase | Placebo
Started | 0 | 88 (Only those participants who completed OL phase, achieved at least a JIA ACR 30 response in OL phase.) | 85 (Only those participants who completed OL phase,achieved at least a JIA ACR 30 response in OL phase.)
Treated | 0 | 88 | 85
Completed | 0 | 61 | 38
Not Completed | 0 | 27 | 47
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Insufficient Clinical Response | 0 | 22 | 44
Not completed — Other | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Medication error without associated AEs | 0 | 1 | 0
Not completed — Withdrawal By Parent/Guardian | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The open-label phase full analysis set (OLFAS) consisted of all participants who were enrolled into open-label phase of the study and received at least one dose of study medication in open-label phase.
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 225
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 11.92 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64
  Not Hispanic or Latino | 161
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 196
  More than one race | 0
  Unknown or Not Reported | 24

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Phase: Percentage of Participants With Disease Flare According to Pediatric Rheumatology Collaborative Study Group/Pediatric Rheumatology International Trials Organization (PRCSG/PRINTO) Disease Flare Criteria at Week 44
Description: According to PRCSG/PRINTO, disease flare defined as worsening of >=30 percent(%) in >=3 of 6 variables of JIA core set, with no more than 1 variable improving by >=30%. Six core variables: 1) Number of joints with active arthritis (joint with swelling/in absence of swelling, limited range of motion accompanied by pain/tenderness), 2)Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a Visual Analog Scale[VAS] of 0[no activity] to 10[maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on VAS of 0[very well] to 10[very poor], 5) Childhood Health Assessment Questionnaire- Disability Index (CHAQ-DI): 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score,which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) Erythrocyte Sedimentation Rate(ESR).
Time Frame: Week 44
Population: The Double Blind polyarticular course JIA analysis set (DBJAS) included all participants randomized to the double-blind phase, received at least 1 dose of study medication in the double-blind phase and had polyarticular course JIA.
Measure: Number; unit: percentage of participants
Groups:
- Tofacitinib: Double Blind Phase: Participants who completed open-label phase and achieved at least a JIA ACR 30 response in open label phase, were randomized at Week 18 to receive tofacitinib tablets (for participants >=40 body weight) or oral solution (for participants <40 kg body weight), BID, in double-blind phase for additional 26 weeks (up to Week 44).
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants | 29.17 | 52.86
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; In order to preserve type I error, each endpoint assessed sequentially using gate-keeping or step-down approach where statistical significance was claimed for the second endpoint only if the first endpoint in the sequence meets the requirements for significance; Test type: Superiority; p = 0.0031, Normal approximation to the binomial — Threshold for significance at 0.05 level; Difference in percentage = -23.69, 95% CI 2-sided [-39.41 to -7.97]

2. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 50 Response at Week 44
Description: JIA ACR50 response defined as: >=50% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction); 6) ESR.
Time Frame: Week 44
Population: The DBJAS included all participants randomized to the double-blind phase, received at least 1 dose of study medication in the double-blind phase and had polyarticular course JIA.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants | 66.67 | 47.14
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0166, Normal approximation to the binomial — Threshold for significance at 0.05 level; Difference in percentage = 19.52, 95% CI 2-sided [3.55 to 35.50]

3. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 Response at Week 44
Description: JIA ACR30 response defined as: >=30% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction); 6) ESR.
Time Frame: Week 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants | 70.83 | 47.14
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0031, Normal approximation to the binomial — Threshold for significance at 0.05 level; Difference in percentage = 23.69, 95% CI 2-sided [7.97 to 39.41]

4. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 70 Response at Week 44
Description: JIA ACR70 response defined as: >=70% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction); 6) ESR.
Time Frame: Week 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants | 54.17 | 37.14
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0387, Normal approximation to the binomial — Threshold for significance at 0.05 level; Difference in percentage = 17.02, 95% CI 2-sided [0.88 to 33.17]

5. Secondary Outcome: Double Blind Phase: JIA ACR Core Variable- Change From Double-Blind Baseline in Childhood Health Assessment Questionnaire- Disability Index (CHAQ-DI) Total Score at Week 44
Description: CHAQ is a valid assessment of functional disability, discomfort in participants with rheumatic diseases. It comprises of three indices: Disability and Discomfort, and global assessment of arthritis (overall well-being). CHAQ-DI: as a measure of functional ability, consists of 30 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities-distributed, among a total of 30 items. Each question was rated on a 4-point scale of difficulty in performance ranges from 0 (no difficulty) to 3 (unable to do). To calculate the overall score, the participant must have a domain score in at least 6 of the 8 domains. Scores of 8 domains were averaged to calculate the CHAQ-DI total score which ranges from 0 (no or minimal physical dysfunction) to 3 (very severe physical dysfunction), higher score indicates more disability. Change from double-blind baseline at Week 44 in DI total score is reported.
Time Frame: Baseline, Week 44
Population: The DBJAS included all participants randomized to the double-blind phase, received at least 1 dose of study medication in the double-blind phase and had polyarticular course JIA. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 49 | 33
units on a scale | -0.09 (0.04) | 0.03 (0.04)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; In order to preserve type I error, each endpoint assessed sequentially using gate-keeping or step-down approach where statistical significance was claimed for the second endpoint only if the first endpoint in the sequence meets the requirements for significance. Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.0292, Mixed Model for Repeated Measures (MMRM) — Threshold for significance at 0.05 level; Ls mean difference = -0.12, 95% CI 2-sided [-0.22 to -0.01], Standard Error of Mean 0.05

6. Secondary Outcome: Open-Label Phase: Percentage of Participants With Disease Flare According to Pediatric Rheumatology Collaborative Study Group/Pediatric Rheumatology International Trials Organization (PRCSG/PRINTO) Disease Flare Criteria at Week 2, 4, 8, 12 and 18
Description: According to PRCSG/PRINTO, disease flare defined as worsening of >=30% in >=3 of 6 variables of JIA core set, with no more than 1 variable improving by >=30%. Six core variables were: 1) Number of joints with active arthritis (joint with swelling or in absence of swelling, limited range of motion accompanied by pain/ tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) ESR.
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: The OLJAS included all participants who were enrolled into the open-label phase of the study and received at least one dose of study medication in open-label phase and had polyarticular course JIA. Here, 'number analyzed' (n) signifies participants evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Week 2 | 0.54
  Week 4: number analyzed (Participants) | 183
  Week 4 | 3.83
  Week 8: number analyzed (Participants) | 175
  Week 8 | 5.14
  Week 12: number analyzed (Participants) | 166
  Week 12 | 7.23
  Week 18: number analyzed (Participants) | 154
  Week 18 | 8.44

7. Secondary Outcome: Double Blind Phase: Percentage of Participants With Disease Flare According to PRCSG/PRINTO Disease Flare Criteria at Week 20, 24, 28, 32, 36 and 40
Description: According to PRCSG/PRINTO, disease flare defined as worsening of >=30% in >=3 of 6 variables of JIA core set, with no more than 1 variable improving by >=30%. Six core variables were: 1) Number of joints with active arthritis (joint with swelling or in absence of swelling, limited range of motion accompanied by pain/ tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction); 6) ESR.
Time Frame: Weeks 20, 24, 28, 32, 36 and 40
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Week 20 | 9.72 | 11.43
  Week 24 | 12.50 | 31.43
  Week 28 | 18.06 | 37.14
  Week 32 | 23.61 | 45.71
  Week 36 | 25.00 | 48.57
  Week 40 | 27.78 | 52.86
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 20; Test type: Superiority; p = 0.7410, Normal approximation to the binomial; Difference in percentage = -1.71, 95% CI 2-sided [-11.82 to 8.41]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 24; Test type: Superiority; p = 0.0052, Normal approximation to the binomial; Difference in percentage = -18.93, 95% CI 2-sided [-32.22 to -5.64]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 28; Test type: Superiority; p = 0.0093, Normal approximation to the binomial; Difference in percentage = -19.09, 95% CI 2-sided [-33.48 to -4.70]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 32; Test type: Superiority; p = 0.0045, Normal approximation to the binomial; Difference in percentage = -22.10, 95% CI 2-sided [-37.35 to -6.86]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 36; Test type: Superiority; p = 0.0027, Normal approximation to the binomial; Difference in percentage = -23.57, 95% CI 2-sided [-38.97 to -8.17]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 40; Test type: Superiority; p = 0.0016, Normal approximation to the binomial; Difference in percentage = -25.08, 95% CI 2-sided [-40.69 to -9.47]

8. Secondary Outcome: Open-Label Phase: Time to Disease Flare
Description: Time to disease flare:time (in days) from first dose of study drug until the day of disease flare in open-label phase. According to PRCSG/PRINTO, disease flare: worsening of >=30% in >=3 of 6 variables of JIA core set, with no more than 1 variable improving by >=30%. 6 core variables were: 1) Number of joints with active arthritis (joint with swelling or in absence of swelling, limited range of motion accompanied by pain/ tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) ESR.
Time Frame: Day 1 up to week 18
Population: The OLJAS included all participants who were enrolled into the open-label phase of the study and received at least one dose of study medication in open-label phase and had polyarticular course JIA.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
days | NA [NA to NA] — Median, upper and lower limits of 95% CI was not estimable due to small number of participants with the event.

9. Secondary Outcome: Double Blind Phase: Time to Disease Flare
Description: Time to disease flare: time (in days) from first dose of study drug until the day of disease flare in double blind phase. According to PRCSG/PRINTO, disease flare: worsening of >=30% in >=3 of 6 variables of JIA core set, with no more than 1 variable improving by >=30%. 6 core variables were: 1) Number of joints with active arthritis (joint with swelling or in absence of swelling, limited range of motion accompanied by pain/ tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) ESR.
Time Frame: Day 1 of Week 19 up to week 44
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
days | NA [NA to NA] — Median, upper and lower limits of 95% CI was not estimable due to small number of participants with the event. | 155.0 [86.0 to NA] — Upper limit of 95% CI was not estimable due to small number of participants with the event.

10. Secondary Outcome: Open-Label Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 Response at Weeks 2, 4, 8, 12 and 18
Description: as for outcome 3
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: The OLJAS included all participants who were enrolled into the open-label phase of the study and received at least one dose of study medication in open-label phase and had polyarticular course JIA. Here, "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Week 2 | 45.11
  Week 4: number analyzed (Participants) | 183
  Week 4 | 68.31
  Week 8: number analyzed (Participants) | 177
  Week 8 | 79.66
  Week 12: number analyzed (Participants) | 167
  Week 12 | 85.63
  Week 18: number analyzed (Participants) | 154
  Week 18 | 92.21

11. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 Response at Double Blind Baseline, Weeks 20, 24, 28, 32, 36 and 40
Description: as for outcome 3
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36 and 40
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 100.00 | 100.00
  Week 20 | 88.89 | 82.86
  Week 24 | 86.11 | 68.57
  Week 28 | 80.56 | 61.43
  Week 32 | 76.39 | 52.86
  Week 36 | 73.61 | 48.57
  Week 40 | 70.83 | 47.14
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 20; Test type: Superiority; p = 0.3010, Normal approximation to the binomial; Difference in percentage = 6.03, 95% CI 2-sided [-5.40 to 17.46]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 24; Test type: Superiority; p = 0.0108, Normal approximation to the binomial; Difference in percentage = 17.54, 95% CI 2-sided [4.05 to 31.03]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 28; Test type: Superiority; p = 0.0103, Normal approximation to the binomial; Difference in percentage = 19.13, 95% CI 2-sided [4.51 to 33.74]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 32; Test type: Superiority; p = 0.0025, Normal approximation to the binomial; Difference in percentage = 23.53, 95% CI 2-sided [8.27 to 38.80]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 36; Test type: Superiority; p = 0.0016, Normal approximation to the binomial; Difference in percentage = 25.04, 95% CI 2-sided [9.52 to 40.56]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; at Week 40; Test type: Superiority; p = 0.0031, Normal approximation to the binomial; Difference in percentage = 23.69, 95% CI 2-sided [7.97 to 39.41]

12. Secondary Outcome: Open-Label Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 50 Response at Weeks 2, 4, 8, 12 and 18
Description: JIA ACR50 response defined as: >=50% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) ESR.
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Week 2 | 20.11
  Week 4: number analyzed (Participants) | 183
  Week 4 | 44.81
  Week 8: number analyzed (Participants) | 177
  Week 8 | 62.71
  Week 12: number analyzed (Participants) | 167
  Week 12 | 71.86
  Week 18: number analyzed (Participants) | 154
  Week 18 | 83.77

13. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 50 Response at Double Blind Baseline, Weeks 20, 24, 28, 32, 36 and 40
Description: as for outcome 2
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36 and 40
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 90.28 | 91.43
  Week 20 | 81.94 | 74.29
  Week 24 | 80.56 | 58.57
  Week 28 | 73.61 | 55.71
  Week 32 | 69.44 | 44.29
  Week 36 | 68.06 | 47.14
  Week 40 | 68.06 | 45.71
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Double Blind Baseline (Week 18); Test type: Superiority; p = 0.8119, Normal approximation for binomial; Difference in percentage = -1.15, 95% CI 2-sided [-10.63 to 8.33]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Test type: Superiority; p = 0.2682, Normal approximation for binomial; Difference in percentage = 7.66, 95% CI 2-sided [-5.90 to 21.21]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24; Test type: Superiority; p = 0.0034, Normal approximation for binomial; Difference in percentage = 21.98, 95% CI 2-sided [7.26 to 36.71]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28; Test type: Superiority; p = 0.0233, Normal approximation for binomial; Difference in percentage = 17.90, 95% CI 2-sided [2.44 to 33.36]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32; Test type: Superiority; p = 0.0018, Normal approximation for binomial; Difference in percentage = 25.16, 95% CI 2-sided [9.39 to 40.93]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36; Test type: Superiority; p = 0.0099, Normal approximation for binomial; Difference in percentage = 20.91, 95% CI 2-sided [5.01 to 36.81]
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40; Test type: Superiority; p = 0.0058, Normal approximation for binomial; Difference in percentage = 22.34, 95% CI 2-sided [6.46 to 38.22]

14. Secondary Outcome: Open-Label Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 70 Response at Weeks 2, 4, 8, 12 and 18
Description: JIA ACR70 response defined as: >=70% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) ESR.
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Week 2 | 7.61
  Week 4: number analyzed (Participants) | 183
  Week 4 | 16.94
  Week 8: number analyzed (Participants) | 177
  Week 8 | 36.16
  Week 12: number analyzed (Participants) | 167
  Week 12 | 46.71
  Week 18: number analyzed (Participants) | 154
  Week 18 | 61.04

15. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 70 Response at Double Blind Baseline (Week 18),Week 20, 24, 28, 32, 36 and 40
Description: as for outcome 4
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36 and 40
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 68.06 | 64.29
  Week 20 | 58.33 | 55.71
  Week 24 | 58.33 | 44.29
  Week 28 | 54.17 | 47.14
  Week 32 | 56.94 | 38.57
  Week 36 | 54.17 | 34.29
  Week 40 | 54.17 | 34.29
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Double Blind Baseline (Week 18); Test type: Superiority; p = 0.6348, Normal approximation to the binomial; Difference in percentage = 3.77, 95% CI 2-sided [-11.79 to 19.33]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Test type: Superiority; p = 0.7525, Normal approximation to the binomial; Difference in percentage = 2.62, 95% CI 2-sided [-13.66 to 18.90]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24; Test type: Superiority; p = 0.0908, Normal approximation to the binomial; Difference in percentage = 14.05, 95% CI 2-sided [-2.23 to 30.33]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28; Test type: Superiority; p = 0.4026, Normal approximation to the binomial; Difference in percentage = 7.02, 95% CI 2-sided [-9.38 to 23.43]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32; Test type: Superiority; p = 0.0258, Normal approximation to the binomial; Difference in percentage = 18.37, 95% CI 2-sided [2.22 to 34.52]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36; Test type: Superiority; p = 0.0149, Normal approximation to the binomial; Difference in percentage = 19.88, 95% CI 2-sided [3.88 to 35.88]
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40; Test type: Superiority; p = 0.0149, Normal approximation to the binomial; Difference in percentage = 19.88, 95% CI 2-sided [3.88 to 35.88]

16. Secondary Outcome: Open-Label Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 90 Response at Week 2, 4, 8, 12 and 18
Description: JIA ACR90 response defined as: >=90% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction); 6) ESR.
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: The OLJAS included all participants who were enrolled into the open-label phase of the study and received at least one dose of study medication in open-label phase and had polyarticular course JIA. Here "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Week 2 | 0
  Week 4: number analyzed (Participants) | 183
  Week 4 | 3.83
  Week 8: number analyzed (Participants) | 177
  Week 8 | 11.30
  Week 12: number analyzed (Participants) | 167
  Week 12 | 20.96
  Week 18: number analyzed (Participants) | 154
  Week 18 | 33.12

17. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 90 Response at Double Blind Baseline (Week 18), Week 20, 24, 28, 32, 36, 40 and 44
Description: JIA ACR90 response defined as: >=90% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) ESR.
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 33.33 | 38.57
  Week 20 | 34.72 | 25.71
  Week 24 | 37.50 | 28.57
  Week 28 | 36.11 | 27.14
  Week 32 | 38.89 | 22.86
  Week 36 | 38.89 | 20.00
  Week 40 | 34.72 | 22.86
  Week 44 | 34.72 | 21.43
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Double Blind Baseline (Week 18); Test type: Superiority; p = 0.5150, Normal approximation to the binomial; Difference in percentage = -5.24, 95% CI 2-sided [-21.00 to 10.53]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Test type: Superiority; p = 0.2400, Normal approximation to the binomial; Difference in percentage = 9.01, 95% CI [-6.02 to 24.03]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24; Test type: Superiority; p = 0.2557, Normal approximation to the binomial; Difference in percentage = 8.93, 95% CI 2-sided [-6.47 to 24.33]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28; Test type: Superiority; p = 0.2481, Normal approximation to the binomial; Difference in percentage = 8.97, 95% CI 2-sided [-6.25 to 24.19]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32; Test type: Superiority; p = 0.0356, Normal approximation to the binomial; Difference in percentage = 16.03, 95% CI 2-sided [1.08 to 30.98]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36; Test type: Superiority; p = 0.0115, Normal approximation to the binomial; Difference in percentage = 18.89, 95% CI 2-sided [4.24 to 33.54]
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40; Test type: Superiority; p = 0.1150, Normal approximation to the binomial; Difference in percentage = 11.87, 95% CI 2-sided [-2.89 to 26.62]
Statistical Analysis 8: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 44; Test type: Superiority; p = 0.0744, Normal approximation to the binomial; Difference in percentage = 13.29, 95% CI 2-sided [-1.31 to 27.90]

18. Secondary Outcome: Open-Label Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 100 Response at Week 2, 4, 8, 12 and 18
Description: JIA ACR100 response defined as: >=100% improvement in 3 out of 6 JIA core set variables with no more than 1 out of 6 JIA core set variables worsened by >=30%. Six core variables: 1) Number of joints with active arthritis (defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 2) Number of joints with limited range of motion, 3) Physician global evaluation of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 4) Parent/legal guardian/participant global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor], 5) CHAQ-DI: 30 questions in 8 domains, each question answered on scale of 0=without difficulty to 3=unable to do; scores of each domain were averaged to derive total CHAQ-DI score, which ranges from 0 (minimum dysfunction) to 3 (most severe dysfunction);6) ESR.
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Week 2 | 0.0
  Week 4: number analyzed (Participants) | 183
  Week 4 | 2.19
  Week 8: number analyzed (Participants) | 177
  Week 8 | 8.47
  Week 12: number analyzed (Participants) | 167
  Week 12 | 14.37
  Week 18: number analyzed (Participants) | 154
  Week 18 | 21.43

19. Secondary Outcome: Double Blind Phase: Percentage of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 100 Response at Double Blind Baseline (Week 18), Week 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 18
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 15.28 | 31.43
  Week 20 | 27.78 | 17.14
  Week 24 | 27.78 | 24.29
  Week 28 | 26.39 | 24.29
  Week 32 | 27.78 | 21.43
  Week 36 | 30.56 | 18.57
  Week 40 | 29.17 | 20.00
  Week 44 | 29.17 | 17.14
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Double Blind Baseline (Week 18); Test type: Superiority; p = 0.0207, Normal approximation to the binomial; Difference in percentage = -16.15, 95% CI 2-sided [-29.84 to -2.46]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Test type: Superiority; p = 0.1254, Normal approximation to the binomial; Difference in percentage = 10.63, 95% CI 2-sided [-2.97 to 24.24]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24; Test type: Superiority; p = 0.6350, Normal approximation to the binomial; Difference in percentage = 3.49, 95% CI 2-sided [-10.93 to 17.91]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28; Test type: Superiority; p = 0.7732, Normal approximation to the binomial; Difference in percentage = 2.10, 95% CI 2-sided [-12.20 to 16.41]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32; Test type: Superiority; p = 0.3782, Normal approximation to the binomial; Difference in percentage = 6.35, 95% CI 2-sided [-7.77 to 20.47]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36; Test type: Superiority; p = 0.0936, Normal approximation to the binomial; Difference in percentage = 11.98, 95% CI 2-sided [-2.02 to 25.99]
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40; Test type: Superiority; p = 0.2017, Normal approximation to the binomial; Difference in percentage = 9.17, 95% CI 2-sided [-4.91 to 23.24]
Statistical Analysis 8: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 44; Test type: Superiority; p = 0.0858, Normal approximation to the binomial; Difference in percentage = 12.02, 95% CI 2-sided [-1.69 to 25.74]

20. Secondary Outcome: Open Label Phase: Change From Baseline in Juvenile Arthritis Disease Activity Score 27 (JADAS-27) C-Reactive Protein (CRP) Score at Weeks 2, 4, 8, 12 and 18
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 CRP score was derived from four components; 1) Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 2) Parent/legal guardian/subject global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor]), 3) Number of joints with active disease(defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 4) CRP (measured in milligram per liter [mg/L] and value normalized to 0 to 10 scale). The overall JADAS-27 score ranges from 0-57. A higher score indicates more disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
score on scale
  Week 2: number analyzed (Participants) | 181
  Week 2 | -6.35 (5.44)
  Week 4: number analyzed (Participants) | 180
  Week 4 | -9.89 (6.54)
  Week 8: number analyzed (Participants) | 175
  Week 8 | -12.47 (7.51)
  Week 12: number analyzed (Participants) | 163
  Week 12 | -14.33 (6.96)
  Week 18: number analyzed (Participants) | 153
  Week 18 | -15.80 (7.12)

21. Secondary Outcome: Double Blind Phase: Change From Double-Blind Baseline in Juvenile Arthritis Disease Activity Score (JADAS) 27 C-Reactive Protein (CRP) Score at Week 20, 24, 28, 32, 36, 40 and 44
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 CRP score was derived from four components; 1) Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 2) Parent/legal guardian/subject global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor]), 3) Number of joints with active disease(defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 4) CRP (measured in mg/L and value normalized to 0 to 10 scale). The overall JADAS-27 score ranges from 0-57. A higher score indicates more disease activity.
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: The DBJAS included all participants randomized to the double-blind phase, received at least 1 dose of study medication in the double-blind phase and had polyarticular course JIA. Here, "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
score on scale
  Week 20: number analyzed (Participants) | 70 | 69
  Week 20 | 0.27 (0.64) | 2.33 (0.64)
  Week 24: number analyzed (Participants) | 65 | 59
  Week 24 | 0.83 (0.95) | 4.46 (0.97)
  Week 28: number analyzed (Participants) | 63 | 47
  Week 28 | 0.51 (0.91) | 4.36 (0.97)
  Week 32: number analyzed (Participants) | 59 | 43
  Week 32 | 0.16 (0.73) | 3.46 (0.81)
  Week 36: number analyzed (Participants) | 54 | 36
  Week 36 | 0.34 (1.09) | 6.55 (1.22)
  Week 40: number analyzed (Participants) | 53 | 34
  Week 40 | 0.85 (1.13) | 7.11 (1.26)
  Week 44: number analyzed (Participants) | 49 | 32
  Week 44 | 0.03 (0.91) | 4.39 (1.00)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.0088, MMRM; LS mean difference = -2.07, 95% CI 2-sided [-3.60 to -0.53], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24: Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.0054, MMRM; LS mean difference = -3.64, 95% CI 2-sided [-6.17 to -1.10], Standard Error of Mean 1.28
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28: Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.0039, MMRM; LS mean difference = -3.85, 95% CI 2-sided [-6.38 to -1.32], Standard Error of Mean 1.25
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32: Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.0022, MMRM; LS mean difference = -3.30, 95% CI 2-sided [-5.30 to -1.29], Standard Error of Mean 0.98
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36: Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.0005, MMRM; LS mean difference = -6.21, 95% CI 2-sided [-9.42 to -3.00], Standard Error of Mean 1.57
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40: Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.0006, MMRM; LS mean difference = -6.26, 95% CI 2-sided [-9.60 to -2.92], Standard Error of Mean 1.63
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 44: Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.0027, MMRM; LS mean difference = -4.36, 95% CI 2-sided [-7.02 to -1.71], Standard Error of Mean 1.27

22. Secondary Outcome: Open Label Phase: Change From Baseline in JADAS-27 Erythrocyte Sedimentation Rate (ESR) Score at Week 2, 4, 8, 12 and 18
Description: JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 ESR score was derived from four components; 1) Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 2) Parent/legal guardian/subject global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor]), 3) Number of joints with active disease (maximum of 27 and defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 4) ESR. The overall JADAS-27 score ranges from 0-57. A higher score indicates more disease activity.
Time Frame: Baseline, weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
score on scale
  Week 2: number analyzed (Participants) | 180
  Week 2 | -6.38 (5.52)
  Week 4: number analyzed (Participants) | 180
  Week 4 | -10.14 (6.63)
  Week 8: number analyzed (Participants) | 174
  Week 8 | -12.60 (7.60)
  Week 12: number analyzed (Participants) | 165
  Week 12 | -14.54 (6.90)
  Week 18: number analyzed (Participants) | 154
  Week 18 | -15.94 (7.17)

23. Secondary Outcome: Double Blind Phase: Change From Double-Blind Baseline in JADAS-27 Erythrocyte Sedimentation Rate (ESR) Score at Weeks 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 22
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
score on scale
  Week 20: number analyzed (Participants) | 71 | 70
  Week 20 | 0.62 (0.62) | 2.45 (0.62)
  Week 24: number analyzed (Participants) | 66 | 60
  Week 24 | 0.92 (0.90) | 4.33 (0.92)
  Week 28: number analyzed (Participants) | 63 | 49
  Week 28 | 0.64 (0.86) | 4.22 (0.90)
  Week 32: number analyzed (Participants) | 59 | 45
  Week 32 | 0.26 (0.75) | 3.67 (0.81)
  Week 36: number analyzed (Participants) | 55 | 37
  Week 36 | 0.60 (1.06) | 6.26 (1.17)
  Week 40: number analyzed (Participants) | 53 | 35
  Week 40 | 0.73 (1.05) | 6.35 (1.15)
  Week 44: number analyzed (Participants) | 49 | 33
  Week 44 | 0.09 (0.91) | 4.50 (0.97)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20: Analysis was based on Mixed Model for Repeated Measures (MMRM) with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.0172, MMRM; LS Mean Difference = -1.83, 95% CI 2-sided [-3.32 to -0.33], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; p = 0.0057, MMRM; LS Mean Difference = -3.41, 95% CI 2-sided [-5.81 to -1.01], Standard Error of Mean 1.21
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; p = 0.0038, MMRM; LS Mean Difference = -3.58, 95% CI 2-sided [-5.94 to -1.23], Standard Error of Mean 1.16
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority; p = 0.0020, MMRM; LS Mean Difference = -3.41, 95% CI 2-sided [-5.47 to -1.36], Standard Error of Mean 1.01
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority; p = 0.0007, MMRM; LS Mean Difference = -5.66, 95% CI 2-sided [-8.74 to -2.57], Standard Error of Mean 1.52
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority; p = 0.0007, MMRM; LS Mean Difference = -5.62, 95% CI 2-sided [-8.66 to -2.58], Standard Error of Mean 1.49
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 44:Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.0018, MMRM; LS Mean Difference = -4.41, 95% CI 2-sided [-6.99 to -1.82], Standard Error of Mean 1.25

24. Secondary Outcome: Open-Label Phase: Percentage of Participants With JADAS-27 CRP Minimum Disease Activity at Weeks 2, 4, 8, 12 and 18
Description: Minimum Disease Activity is defined by a JADAS-27 CRP score less than or equal to 3.8 for participants with polyarthritis, and less than or equal to 2 for participants with oligoarthritis. JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 CRP score was derived from four components; 1) Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 2) Parent/legal guardian/subject global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor]), 3) Number of joints with active disease(maximum of 27 defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 4) CRP (measured in milligram per liter [mg/L] and value normalized to 0 to 10 scale). The overall JADAS-27 score ranges from 0-57. A higher score indicates more disease activity.
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Baseline | 0
  Week 2: number analyzed (Participants) | 183
  Week 2 | 2.19
  Week 4: number analyzed (Participants) | 183
  Week 4 | 9.29
  Week 8: number analyzed (Participants) | 176
  Week 8 | 20.45
  Week 12: number analyzed (Participants) | 165
  Week 12 | 29.09
  Week 18: number analyzed (Participants) | 154
  Week 18 | 44.16

25. Secondary Outcome: Double Blind Phase: Percentage of Participants With JADAS-27 CRP Minimum Disease Activity at Double Blind Baseline (Week 18), Week 20, 24, 28, 32, 36, 40 and 44
Description: Minimum Disease Activity is defined by a JADAS-27 CRP score less than or equal to 3.8 for participants with polyarthritis, and less than or equal to 2 for participants with oligoarthritis. JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 CRP score was derived from four components; 1) Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 2) Parent/legal guardian/subject global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor]), 3) Number of joints with active disease (maximum of 27 and defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 4) CRP (measured in milligram per liter [mg/L] and value normalized to 0 to 10 scale). The overall JADAS-27 score ranges from 0-57. A higher score indicates more disease activity.
Time Frame: Double Blind Baseline (Week 18), Week 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 48.61 | 47.14
  Week 20 | 45.83 | 35.71
  Week 24 | 47.22 | 34.29
  Week 28 | 47.22 | 35.71
  Week 32 | 40.28 | 32.86
  Week 36 | 44.44 | 30.00
  Week 40 | 45.83 | 31.43
  Week 44 | 47.22 | 32.86
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Double Blind Baseline (Week 18); Test type: Superiority; p = 0.8610, Normal approximation to the binomial; Difference in percentage = 1.47, 95% CI 2-sided [-14.96 to 17.90]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Test type: Superiority; p = 0.2173, Normal approximation to the binomial; Difference in percentage = 10.12, 95% CI 2-sided [-5.96 to 26.20]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24; Test type: Superiority; p = 0.1135, Normal approximation to the binomial; Difference in percentage = 12.94, 95% CI 2-sided [-3.08 to 28.96]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28; Test type: Superiority; p = 0.1610, Normal approximation to the binomial; Difference in percentage = 11.51, 95% CI 2-sided [-4.58 to 27.60]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32; Test type: Superiority; p = 0.3571, Normal approximation to the binomial; Difference in percentage = 7.42, 95% CI 2-sided [-8.37 to 23.21]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36; Test type: Superiority; p = 0.0716, Normal approximation to the binomial; Difference in percentage = 14.44, 95% CI 2-sided [-1.27 to 30.16]
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40; Test type: Superiority; p = 0.0746, Normal approximation to the binomial; Difference in percentage = 14.40, 95% CI 2-sided [-1.43 to 30.24]
Statistical Analysis 8: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 44; Test type: Superiority; p = 0.0773, Normal approximation to the binomial; Difference in percentage = 14.37, 95% CI 2-sided [-1.57 to 30.30]

26. Secondary Outcome: Open-Label Phase: Percentage of Participants With JADAS-27 CRP Inactive Disease Activity at Week 2, 4, 8, 12 and 18
Description: JADAS-27 inactive disease is defined by a JADAS score less than or equal to 1. JADAS-27 Inactive Disease cutoff values are defined as: 1) Polyarthritis: Inactive Disease: <=1 and 2) Oligoarthritis (<4 active joints): Inactive Disease: <=1. JADAS-27 is a validated composite disease activity measure for JIA. JADAS-27 CRP score was derived from four components; 1) Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]), 2) Parent/legal guardian/subject global assessment of overall well-being (assessed on a VAS of 0 [very well] to 10 [very poor]), 3) Number of joints with active disease (maximum of 27 and defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness), 4) CRP (measured in milligram per liter [mg/L] and value normalized to 0 to 10 scale). The overall JADAS-27 score ranges from 0-57. A higher score indicates more disease activity.
Time Frame: Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
percentage of participants
  Week 2: number analyzed (Participants) | 183
  Week 2 | 0
  Week 4: number analyzed (Participants) | 183
  Week 4 | 0
  Week 8: number analyzed (Participants) | 176
  Week 8 | 2.84
  Week 12: number analyzed (Participants) | 165
  Week 12 | 3.64
  Week 18: number analyzed (Participants) | 154
  Week 18 | 7.79

27. Secondary Outcome: Double Blind Phase: Percentage of Participants With JADAS-27 CRP Inactive Disease Activity at Double Blind Baseline (Week 18), Week 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 26
Time Frame: Double Blind Baseline (Week 18), Week 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 6.94 | 10.00
  Week 20 | 9.72 | 2.86
  Week 24 | 12.50 | 5.71
  Week 28 | 9.72 | 7.14
  Week 32 | 11.11 | 5.71
  Week 36 | 16.67 | 7.14
  Week 40 | 18.06 | 7.14
  Week 44 | 18.06 | 10.00
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Double Blind Baseline (Week 18); Test type: Superiority; p = 0.5131, Normal approximation to the binomial; Difference in percentage = -3.06, 95% CI 2-sided [-12.21 to 6.10]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Test type: Superiority; p = 0.0876, Normal approximation to the binomial; Difference in percentage = 6.87, 95% CI 2-sided [-1.01 to 14.74]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24; Test type: Superiority; p = 0.1561, Normal approximation to the binomial; Difference in percentage = 6.79, 95% CI 2-sided [-2.59 to 16.16]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28; Test type: Superiority; p = 0.5795, Normal approximation to the binomial; Difference in percentage = 2.58, 95% CI 2-sided [-6.54 to 11.70]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32; Test type: Superiority; p = 0.2435, Normal approximation to the binomial; Difference in percentage = 5.40, 95% CI 2-sided [-3.67 to 14.47]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36; Test type: Superiority; p = 0.0758, Normal approximation to the binomial; Difference in percentage = 9.52, 95% CI 2-sided [-0.99 to 20.04]
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40; Test type: Superiority; p = 0.0464, Normal approximation to the binomial; Difference in percentage = 10.91, 95% CI 2-sided [0.17 to 21.65]
Statistical Analysis 8: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 44; Test type: Superiority; p = 0.1634, Normal approximation to the binomial; Difference in percentage = 8.06, 95% CI 2-sided [-3.27 to 19.38]

28. Secondary Outcome: Double Blind Phase: Percentage of Participants With JIA ACR Inactive Disease at Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Description: JIA ACR Inactive Disease criteria included: No joints with active arthritis, No fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to sJIA, No active uveitis (as defined by the Standardized Uveitis Nomenclature (SUN) Working Group), Normal ESR (within normal limits of the method used where tested) or, if elevated, not attributable to JIA, Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]) score of 'best possible' (score of "0") on the scale used, morning stiffness of <=15 minutes.
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants
  Double Blind Baseline (Week 18) | 9.72 | 27.14
  Week 20 | 15.28 | 15.71
  Week 24 | 20.83 | 21.43
  Week 28 | 19.44 | 18.57
  Week 32 | 22.22 | 20.00
  Week 36 | 26.39 | 17.14
  Week 40 | 26.39 | 14.29
  Week 44 | 26.39 | 17.14
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Double Blind baseline (Week 18); Test type: Superiority; p = 0.0062, Normal approximation to the binomial; Difference in percentage = -17.42, 95% CI 2-sided [-29.88 to -4.96]
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20; Test type: Superiority; p = 0.9427, Normal approximation to the binomial; Difference in percentage = -0.44, 95% CI 2-sided [-12.34 to 11.47]
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 24; Test type: Superiority; p = 0.9308, Normal approximation to the binomial; Difference in percentage = -0.60, 95% CI 2-sided [-14.03 to 12.84]
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 28; Test type: Superiority; p = 0.8945, Normal approximation to the binomial; Difference in percentage = 0.87, 95% CI 2-sided [-12.03 to 13.78]
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 32; Test type: Superiority; p = 0.7455, Normal approximation to the binomial; Difference in percentage = 2.22, 95% CI 2-sided [-11.20 to 15.64]
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 36; Test type: Superiority; p = 0.1787, Normal approximation to the binomial; Difference in percentage = 9.25, 95% CI 2-sided [-4.23 to 22.72]
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 40; Test type: Superiority; p = 0.0695, Normal approximation to the binomial; Difference in percentage = 12.10, 95% CI 2-sided [-0.97 to 25.17]
Statistical Analysis 8: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 44; Test type: Superiority; p = 0.1787, Normal approximation to the binomial; Difference in percentage = 9.25, 95% CI 2-sided [-4.23 to 22.72]

29. Secondary Outcome: Double Blind Phase: Percentage of Participants With Presence of JIA ACR Clinical Remission
Description: JIA ACR Clinical Remission Criteria included: Clinical inactive disease for 6 months continuously while on medications for JIA. Clinical Inactive Disease criteria included: No joints with active arthritis, No fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to sJIA, No active uveitis (as defined by the SUN Working Group), Normal ESR (within normal limits of the method used where tested) or, if elevated, not attributable to JIA, Physician global assessment of disease activity (assessed on a VAS of 0 [no activity] to 10 [maximum activity]) score of 'best possible' (score of "0") on the scale used, morning stiffness of less than or equal to (<=) 15 minutes.
Time Frame: From Week 18 in double blind phase up to Week 44
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
percentage of participants | 4.17 | 4.29
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Test type: Superiority; p = 0.9719, Normal approximation to the binomial; Difference in percentage = -0.12, 95% CI 2-sided [-6.74 to 6.50]

30. Secondary Outcome: Open Label Phase: JIA ACR Core Variable- Change From Baseline in Number of Joints With Active Arthritis at Week 2, 4, 8, 12 and 18
Description: Number of joints with active arthritis defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness. The score range of the number of joints is from 0-71.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: joints with active arthritis
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
joints with active arthritis
  Week 2: number analyzed (Participants) | 183
  Week 2 | -4.54 (5.33)
  Week 4: number analyzed (Participants) | 181
  Week 4 | -7.21 (6.36)
  Week 8: number analyzed (Participants) | 175
  Week 8 | -8.62 (7.04)
  Week 12: number analyzed (Participants) | 166
  Week 12 | -9.76 (6.76)
  Week 18: number analyzed (Participants) | 154
  Week 18 | -10.29 (6.79)

31. Secondary Outcome: Double Blind Phase: JIA ACR Core Variable- Change From Double-Blind Baseline in Number of Joints With Active Arthritis at Weeks 20, 24, 28, 32, 36, 40 and 44
Description: Number of joints with active arthritis defined as joint with swelling or, in absence of swelling, limited range of motion accompanied by either pain on motion or tenderness. Number of joints ranged from 0 to 71.
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: joints with active arthritis
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
joints with active arthritis
  Week 20: number analyzed (Participants) | 71 | 70
  Week 20 | 0.21 (0.48) | 1.07 (0.49)
  Week 24: number analyzed (Participants) | 66 | 60
  Week 24 | 0.69 (0.71) | 2.11 (0.72)
  Week 28: number analyzed (Participants) | 63 | 50
  Week 28 | 0.46 (0.61) | 2.13 (0.64)
  Week 32: number analyzed (Participants) | 59 | 45
  Week 32 | 0.19 (0.48) | 1.36 (0.51)
  Week 36: number analyzed (Participants) | 55 | 37
  Week 36 | 0.52 (0.85) | 4.50 (0.92)
  Week 40: number analyzed (Participants) | 53 | 35
  Week 40 | 0.91 (0.85) | 4.48 (0.93)
  Week 44: number analyzed (Participants) | 49 | 33
  Week 44 | 0.55 (0.74) | 2.79 (0.77)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Week 20: Analysis was based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the double-blind baseline value; Test type: Superiority; p = 0.1595, MMRM; LS Mean Difference = -0.87, 95% CI 2-sided [-2.08 to 0.35], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; p = 0.1421, MMRM; LS Mean difference = -1.42, 95% CI 2-sided [-3.32 to 0.48], Standard Error of Mean 0.96
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; p = 0.0552, MMRM; LS Mean difference = -1.66, 95% CI 2-sided [-3.37 to 0.04], Standard Error of Mean 0.83
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority; p = 0.0822, MMRM; LS Mean difference = -1.17, 95% CI 2-sided [-2.50 to 0.17], Standard Error of Mean 0.63
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority; p = 0.0041, MMRM; LS Mean difference = -3.98, 95% CI 2-sided [-6.53 to -1.43], Standard Error of Mean 1.22
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority; p = 0.0085, MMRM; LS Mean difference = -3.57, 95% CI 2-sided [-6.12 to -1.02], Standard Error of Mean 1.22
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority; p = 0.0384, MMRM; LS Mean difference = -2.24, 95% CI 2-sided [-4.36 to -0.13], Standard Error of Mean 1.03

32. Secondary Outcome: Open Label Phase: JIA ACR Core Variable- Change From Baseline in Number of Joints With Limited Range of Motion at Weeks 2, 4, 8, 12 and 18
Description: The maximum number of joints with limitation of movement was 67 and these were defined as those in the joint assessment with 'limitation of motion'.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: joints with limited range of motion
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
joints with limited range of motion
  Week 2: number analyzed (Participants) | 183
  Week 2 | -2.52 (4.21)
  Week 4: number analyzed (Participants) | 181
  Week 4 | -3.56 (5.68)
  Week 8: number analyzed (Participants) | 175
  Week 8 | -4.53 (5.65)
  Week 12: number analyzed (Participants) | 166
  Week 12 | -5.09 (5.79)
  Week 18: number analyzed (Participants) | 154
  Week 18 | -5.77 (5.82)

33. Secondary Outcome: Double Blind Phase: JIA ACR Core Variable- Change From Double-Blind Baseline in Number of Joints With Limited Range of Motion at Double Blind Baseline (Week 18), Week 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 32
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: joints with limited range of motion
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
joints with limited range of motion
  Week 20: number analyzed (Participants) | 71 | 70
  Week 20 | 0.38 (0.20) | 0.64 (0.19)
  Week 24: number analyzed (Participants) | 66 | 60
  Week 24 | 0.50 (0.28) | 1.19 (0.29)
  Week 28: number analyzed (Participants) | 63 | 50
  Week 28 | 0.68 (0.35) | 1.63 (0.37)
  Week 32: number analyzed (Participants) | 59 | 45
  Week 32 | 0.61 (0.32) | 1.40 (0.34)
  Week 36: number analyzed (Participants) | 55 | 37
  Week 36 | 0.47 (0.31) | 1.48 (0.34)
  Week 40: number analyzed (Participants) | 53 | 35
  Week 40 | 0.41 (0.34) | 1.49 (0.39)
  Week 44: number analyzed (Participants) | 49 | 33
  Week 44 | 0.38 (0.29) | 1.20 (0.34)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.2595, MMRM; LS Mean Difference = -0.26, 95% CI 2-sided [-0.72 to 0.19], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; p = 0.0674, MMRM; LS Mean difference = -0.69, 95% CI 2-sided [-1.42 to 0.05], Standard Error of Mean 0.37
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; p = 0.0580, MMRM; LS Mean difference = -0.95, 95% CI 2-sided [-1.93 to 0.03], Standard Error of Mean 0.49
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority; p = 0.0751, MMRM; LS Mean difference = -0.79, 95% CI 2-sided [-1.67 to 0.08], Standard Error of Mean 0.44
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority; p = 0.0251, MMRM; LS Mean difference = -1.01, 95% CI 2-sided [-1.88 to -0.13], Standard Error of Mean 0.43
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority; p = 0.0331, MMRM; LS Mean difference = -1.08, 95% CI 2-sided [-2.07 to -0.09], Standard Error of Mean 0.49
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority; p = 0.0549, MMRM; LS Mean difference = -0.82, 95% CI 2-sided [-1.66 to 0.02], Standard Error of Mean 0.42

34. Secondary Outcome: Open Label Phase: JIA ACR Core Variable- Change From Baseline in Physician Global Evaluation of Disease Activity at Week 2, 4, 8, 12 and 18
Description: Physician global evaluation of disease activity was measured on a 21-numbered circle VAS ranges from 0 to 10 (in 0.5 increments), with '0' as 'No Activity' and '10' as 'Maximum Activity', higher score indicated more disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
score on scale
  Week 2: number analyzed (Participants) | 183
  Week 2 | -1.81 (1.52)
  Week 4: number analyzed (Participants) | 181
  Week 4 | -2.78 (1.84)
  Week 8: number analyzed (Participants) | 175
  Week 8 | -3.51 (1.83)
  Week 12: number analyzed (Participants) | 166
  Week 12 | -4.04 (1.88)
  Week 18: number analyzed (Participants) | 154
  Week 18 | -4.54 (1.92)

35. Secondary Outcome: Double Blind Phase: JIA ACR Core Variable- Change From Double-Blind Baseline in Physician Global Evaluation of Disease Activity at Weeks 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 34
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
score on scale
  Week 20: number analyzed (Participants) | 71 | 70
  Week 20 | 0.28 (0.20) | 0.82 (0.20)
  Week 24: number analyzed (Participants) | 66 | 60
  Week 24 | 0.24 (0.24) | 1.08 (0.24)
  Week 28: number analyzed (Participants) | 63 | 50
  Week 28 | 0.12 (0.21) | 0.92 (0.92)
  Week 32: number analyzed (Participants) | 59 | 45
  Week 32 | -0.03 (0.20) | 0.86 (0.22)
  Week 36: number analyzed (Participants) | 55 | 37
  Week 36 | 0.14 (0.28) | 1.56 (0.32)
  Week 40: number analyzed (Participants) | 53 | 35
  Week 40 | 0.02 (0.28) | 1.64 (0.32)
  Week 44: number analyzed (Participants) | 49 | 33
  Week 44 | -0.16 (0.29) | 1.42 (0.34)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.0353, MMRM; LS mean difference = -0.54, 95% CI 2-sided [-1.04 to -0.04], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; p = 0.0094, MMRM; LS Mean difference = -0.84, 95% CI 2-sided [-1.47 to -0.21], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; p = 0.0065, MMRM; LS Mean difference = -0.80, 95% CI 2-sided [-1.36 to -0.23], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority; p = 0.0018, MMRM; LS Mean difference = -0.89, 95% CI 2-sided [-1.43 to -0.34], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority; p = 0.0010, MMRM; LS Mean difference = -1.42, 95% CI 2-sided [-2.24 to -0.61], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority; p = 0.0002, MMRM; LS Mean difference = -1.61, 95% CI 2-sided [-2.42 to -0.81], Standard Error of Mean 0.40
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority; p = 0.0007, MMRM; LS Mean difference = -1.58, 95% CI 2-sided [-2.44 to -0.71], Standard Error of Mean 0.43

36. Secondary Outcome: Open Label Phase: JIA ACR Core Variable- Change From Baseline in Parent/Legal Guardian/Participant Global Evaluation of Overall Well-Being at Weeks 2, 4, 8, 12 and 18
Description: The parent/or legal guardian/participant rated the overall well-being on a 21-numbered circle VAS ranges from 0 to 10 (in 0.5 increments), with '0' as 'Very Well' and '10' as 'Very Poorly', higher scores=more disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
score on scale
  Week 2: number analyzed (Participants) | 182
  Week 2 | -0.94 (1.95)
  Week 4: number analyzed (Participants) | 181
  Week 4 | -1.47 (1.92)
  Week 8: number analyzed (Participants) | 175
  Week 8 | -1.90 (2.20)
  Week 12: number analyzed (Participants) | 165
  Week 12 | -2.30 (2.15)
  Week 18: number analyzed (Participants) | 154
  Week 18 | -2.68 (2.33)

37. Secondary Outcome: Double Blind Phase: JIA ACR Core Variable- Change From Double-Blind Baseline in Parent/Legal Guardian/Participant Global Evaluation of Overall Well-Being at Weeks 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 36
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
score on scale
  Week 20: number analyzed (Participants) | 71 | 70
  Week 20 | -0.04 (0.18) | 0.38 (0.18)
  Week 24: number analyzed (Participants) | 66 | 60
  Week 24 | -0.03 (0.22) | 0.91 (0.22)
  Week 28: number analyzed (Participants) | 63 | 49
  Week 28 | -0.11 (0.24) | 0.72 (0.26)
  Week 32: number analyzed (Participants) | 59 | 45
  Week 32 | -0.15 (0.24) | 0.82 (0.26)
  Week 36: number analyzed (Participants) | 55 | 37
  Week 36 | -0.22 (0.21) | 0.31 (0.24)
  Week 40: number analyzed (Participants) | 53 | 35
  Week 40 | -0.24 (0.24) | 0.39 (0.27)
  Week 44: number analyzed (Participants) | 49 | 33
  Week 44 | -0.49 (0.22) | 0.24 (0.24)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.0398, MMRM; LS Mean Difference = -0.42, 95% CI 2-sided [-0.83 to -0.02], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; p = 0.0011, MMRM; LS Mean difference = -0.94, 95% CI 2-sided [-1.49 to -0.39], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; p = 0.0131, MMRM; LS mean difference = -0.82, 95% CI 2-sided [-1.47 to -0.18], Standard Error of Mean 0.32
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority; p = 0.0039, MMRM; LS mean difference = -0.97, 95% CI 2-sided [-1.62 to -0.33], Standard Error of Mean 0.32
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority; p = 0.0711, MMRM; LS mean difference = -0.53, 95% CI 2-sided [-1.10 to 0.05], Standard Error of Mean 0.29
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority; p = 0.0658, MMRM; LS mean difference = -0.63, 95% CI 2-sided [-1.30 to 0.04], Standard Error of Mean 0.34
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority; p = 0.0154, MMRM; LS mean difference = -0.73, 95% CI 2-sided [-1.31 to -0.15], Standard Error of Mean 0.29

38. Secondary Outcome: Open Label Phase: JIA ACR Core Variable- Change From Baseline in Childhood Health Assessment Questionnaire- Disability Index (CHAQ-DI) Total Scores at Weeks 2, 4, 8, 12 and 18
Description: CHAQ is a valid assessment of functional disability, discomfort in participants with rheumatic diseases. It comprises of three indices: Disability and Discomfort, and global assessment of arthritis (overall well-being). CHAQ-DI: as a measure of functional ability, consists of 30 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities-distributed, among a total of 30 items. Each question was rated on a 4-point scale of difficulty in performance ranges from 0 (no difficulty) to 3 (unable to do). To calculate the overall score, the participant must have a domain score in at least 6 of the 8 domains. Scores of 8 domains were averaged to calculate the CHAQ-DI total score which ranges from 0 (no or minimal physical dysfunction) to 3 (very severe physical dysfunction), higher score indicates more disability. Change from baseline at Weeks 2, 4, 8, 12 and 18 in DI total score is reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
score on scale
  Week 2: number analyzed (Participants) | 182
  Week 2 | -0.15 (0.41)
  Week 4: number analyzed (Participants) | 181
  Week 4 | -0.23 (0.42)
  Week 8: number analyzed (Participants) | 175
  Week 8 | -0.36 (0.46)
  Week 12: number analyzed (Participants) | 165
  Week 12 | -0.41 (0.53)
  Week 18: number analyzed (Participants) | 154
  Week 18 | -0.49 (0.57)

39. Secondary Outcome: Double Blind Phase: JIA ACR Core Variable- Change From Double-Blind Baseline in Childhood Health Assessment Questionnaire- Disability Index (CHAQ-DI) Total Scores at Weeks 20, 24, 28, 32, 36, and 40
Description: CHAQ: valid assessment of functional disability, discomfort in participants with rheumatic diseases. It comprises of three indices: Disability and Discomfort, and global assessment of arthritis (overall well-being). CHAQ-DI: as a measure of functional ability, consists of 30 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities-distributed, among a total of 30 items. Each question was rated on a 4-point scale of difficulty in performance ranges from 0 (no difficulty) to 3 (unable to do). To calculate overall score, participant must have a domain score in at least 6 of the 8 domains. Scores of 8 domains were averaged to calculate the CHAQ-DI total score which ranges from 0 (no or minimal physical dysfunction) to 3 (very severe physical dysfunction), higher score indicates more disability. Change from double-blind baseline at Weeks 20, 24, 28, 32, 36, and 40 in DI total score is reported.
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, and 40
Population: as for outcome 21
Measure: Least Squares Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
score on scale
  Week 20: number analyzed (Participants) | 71 | 70
  Week 20 | 0.05 (0.04) | 0.08 (0.04)
  Week 24: number analyzed (Participants) | 66 | 59
  Week 24 | 0.01 (0.03) | 0.08 (0.04)
  Week 28: number analyzed (Participants) | 63 | 49
  Week 28 | -0.01 (0.04) | 0.09 (0.04)
  Week 32: number analyzed (Participants) | 59 | 45
  Week 32 | 0.01 (0.04) | 0.10 (0.05)
  Week 36: number analyzed (Participants) | 55 | 37
  Week 36 | -0.04 (0.04) | 0.08 (0.05)
  Week 40: number analyzed (Participants) | 53 | 35
  Week 40 | -0.05 (0.04) | 0.06 (0.05)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.4777, MMRM; LS Mean Difference = -0.03, 95% CI 2-sided [-0.12 to 0.06], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; p = 0.0779, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-0.16 to 0.01], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; p = 0.0324, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.19 to -0.01], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority; p = 0.1061, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.20 to 0.02], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority; p = 0.0572, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.24 to 0.00], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority; p = 0.0689, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.24 to 0.01], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority; p = 0.0292, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.22 to -0.01], Standard Error of Mean 0.05

40. Secondary Outcome: Open-Label Phase: Change From Baseline in Child Health Questionnaire (CHQ) Responses at Week 4 and Week 18
Description: CHQ: 50-item, 14 subscale (Global health, physical functioning, social limitations: emotional, social limitations: physical, bodily pain, behavior, global behavior, mental health, self-esteem, general health, Change in health, emotional impact on parent, time impact on parent, family activities, family cohesion) parent or legal guardian assessed instrument of child's physical, emotional, social well-being, and relative burden of disease on the parents. Each subscale rated on Likert-type scale: range 0 to 100; higher scores indicate a more positive health status. Two summary scores: Physical Health and Psychosocial Health were weighted composites derived from subscale items using scoring algorithms (transformed scores); range 0 to 100: higher scores indicate more positive health status.
Time Frame: Baseline, Week 4 and Week 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
score on scale
  Week 4: Global health: number analyzed (Participants) | 171
  Week 4: Global health | 13.86 (22.40)
  Week 18: Global health: number analyzed (Participants) | 148
  Week 18: Global health | 21.28 (22.79)
  Week 4: Physical functioning: number analyzed (Participants) | 171
  Week 4: Physical functioning | 11.83 (24.47)
  Week 18: Physical functioning: number analyzed (Participants) | 149
  Week 18: Physical functioning | 21.44 (26.78)
  Week 4: Social limitations: emotional: number analyzed (Participants) | 171
  Week 4: Social limitations: emotional | 8.12 (29.29)
  Week 18: Social limitations: emotional: number analyzed (Participants) | 149
  Week 18: Social limitations: emotional | 14.62 (30.18)
  Week 4: Social limitations: physical: number analyzed (Participants) | 171
  Week 4: Social limitations: physical | 13.45 (31.12)
  Week 18: Social limitations: physical: number analyzed (Participants) | 149
  Week 18: Social limitations: physical | 20.81 (32.53)
  Week 4: Bodily pain: number analyzed (Participants) | 171
  Week 4: Bodily pain | 19.42 (21.14)
  Week 18: Bodily pain: number analyzed (Participants) | 149
  Week 18: Bodily pain | 30.60 (22.79)
  Week 4: Behavior: number analyzed (Participants) | 171
  Week 4: Behavior | 3.06 (12.86)
  Week 18: Behavior: number analyzed (Participants) | 149
  Week 18: Behavior | 5.70 (12.91)
  Week 4: Global behavior: number analyzed (Participants) | 171
  Week 4: Global behavior | 7.40 (23.27)
  Week 18: Global behavior: number analyzed (Participants) | 149
  Week 18: Global behavior | 9.30 (24.97)
  Week 4: Mental health: number analyzed (Participants) | 171
  Week 4: Mental health | 6.43 (15.68)
  Week 18: Mental health: number analyzed (Participants) | 149
  Week 18: Mental health | 6.74 (16.06)
  Week 4: Self esteem: number analyzed (Participants) | 171
  Week 4: Self esteem | 2.42 (19.47)
  Week 18: Self esteem: number analyzed (Participants) | 149
  Week 18: Self esteem | 8.45 (17.35)
  Week 4: General health: number analyzed (Participants) | 171
  Week 4: General health | 4.20 (13.50)
  Week 18: General health: number analyzed (Participants) | 149
  Week 18: General health | 7.02 (14.31)
  Week 4: Change in Health: number analyzed (Participants) | 170
  Week 4: Change in Health | 0.86 (1.20)
  Week 18: Change in Health: number analyzed (Participants) | 149
  Week 18: Change in Health | 1.70 (1.32)
  Week 4: Emotional impact on parent: number analyzed (Participants) | 171
  Week 4: Emotional impact on parent | 9.02 (26.30)
  Week 18: Emotional impact on parent: number analyzed (Participants) | 149
  Week 18: Emotional impact on parent | 15.38 (29.35)
  Week 4: Time impact on parent: number analyzed (Participants) | 171
  Week 4: Time impact on parent | 6.17 (24.64)
  Week 18: Time impact on parent: number analyzed (Participants) | 149
  Week 18: Time impact on parent | 9.99 (23.38)
  Week 4: Family activities: number analyzed (Participants) | 171
  Week 4: Family activities | 5.19 (15.15)
  Week 18: Family activities: number analyzed (Participants) | 149
  Week 18: Family activities | 9.59 (19.63)
  Week 4: Family cohesion: number analyzed (Participants) | 171
  Week 4: Family cohesion | 2.78 (21.80)
  Week 18: Family cohesion: number analyzed (Participants) | 149
  Week 18: Family cohesion | 3.62 (18.81)
  Week 4: Physical Health Summary: number analyzed (Participants) | 171
  Week 4: Physical Health Summary | 8.12 (11.18)
  Week 18: Physical Health Summary: number analyzed (Participants) | 149
  Week 18: Physical Health Summary | 13.36 (12.57)
  Week 4: Psychosocial Health Summary: number analyzed (Participants) | 171
  Week 4: Psychosocial Health Summary | 2.46 (8.13)
  Week 18: Psychosocial Health Summary: number analyzed (Participants) | 149
  Week 18: Psychosocial Health Summary | 4.20 (8.41)

41. Secondary Outcome: Double Blind Phase: Change From Double-Blind Baseline in Child Health Questionnaire (CHQ) Responses at Week 44
Description: as for outcome 40
Time Frame: Double-Blind Baseline (Week 18), Week 44
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
score on a scale
  Global health: number analyzed (Participants) | 49 | 30
  Global health | 5.46 (2.83) | 1.66 (3.72)
  Physical functioning: number analyzed (Participants) | 49 | 31
  Physical functioning | 1.45 (3.16) | -1.82 (3.92)
  Social Limitations: Emotional: number analyzed (Participants) | 49 | 31
  Social Limitations: Emotional | 1.78 (3.53) | -3.69 (4.36)
  Social Limitations: Physical: number analyzed (Participants) | 49 | 30
  Social Limitations: Physical | -3.08 (4.03) | -10.29 (5.04)
  Bodily Pain: number analyzed (Participants) | 49 | 31
  Bodily Pain | 6.34 (3.13) | -1.91 (3.91)
  Behavior: number analyzed (Participants) | 49 | 31
  Behavior | 0.78 (2.09) | 4.20 (2.57)
  Global Behavior: number analyzed (Participants) | 49 | 31
  Global Behavior | -2.61 (2.89) | 1.04 (3.54)
  Mental Health: number analyzed (Participants) | 49 | 31
  Mental Health | 0.41 (2.53) | 3.88 (3.12)
  Self Esteem: number analyzed (Participants) | 49 | 31
  Self Esteem | 1.48 (3.29) | 0.76 (4.07)
  General Health: number analyzed (Participants) | 49 | 31
  General Health | 7.91 (1.84) | 6.14 (2.26)
  Change in Health: number analyzed (Participants) | 49 | 31
  Change in Health | 0.07 (0.10) | 0.09 (0.12)
  Emotional Impact on Parent: number analyzed (Participants) | 49 | 31
  Emotional Impact on Parent | 9.55 (4.32) | 0.58 (5.35)
  Time Impact on Parent: number analyzed (Participants) | 49 | 30
  Time Impact on Parent | -3.83 (2.92) | 2.89 (3.62)
  Family Activities: number analyzed (Participants) | 49 | 31
  Family Activities | 0.01 (2.39) | 8.61 (2.95)
  Family Cohesion: number analyzed (Participants) | 49 | 31
  Family Cohesion | 6.04 (3.18) | 3.45 (3.92)
  Physical Health Summary: number analyzed (Participants) | 49 | 30
  Physical Health Summary | 1.67 (1.48) | -1.81 (1.85)
  Psychosocial Health Summary: number analyzed (Participants) | 49 | 30
  Psychosocial Health Summary | 0.64 (1.22) | 1.39 (1.52)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Global Health: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.3179, MMRM; LS Mean Difference = 3.79, 95% CI 2-sided [-3.72 to 11.31], Standard Error of Mean 3.77
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Physical Functioning: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.4452, MMRM; LS mean difference = 3.28, 95% CI 2-sided [-5.23 to 11.78], Standard Error of Mean 4.27
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Social Limitations: Emotional: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.2539, MMRM; LS mean difference = 5.47, 95% CI 2-sided [-4.01 to 14.95], Standard Error of Mean 4.76
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Social Limitations: Physical Subscale: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.1981, MMRM; LS mean difference = 7.22, 95% CI 2-sided [-3.86 to 18.30], Standard Error of Mean 5.56
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase; Bodily Pain: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.0620, MMRM; LS mean difference = 8.26, 95% CI 2-sided [-0.43 to 16.94], Standard Error of Mean 4.36
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Behavior: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.2291, MMRM; LS mean difference = -3.43, 95% CI 2-sided [-9.06 to 2.20], Standard Error of Mean 2.83
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Global Behavior: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.3530, MMRM; LS mean difference = -3.65, 95% CI 2-sided [-11.43 to 4.13], Standard Error of Mean 3.90
Statistical Analysis 8: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Mental Health: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.3114, MMRM; LS mean difference = -3.47, 95% CI 2-sided [-10.26 to 3.32], Standard Error of Mean 3.41
Statistical Analysis 9: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Self Esteem: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.8736, MMRM; LS mean difference = 0.71, 95% CI 2-sided [-8.18 to 9.61], Standard Error of Mean 4.46
Statistical Analysis 10: Comparison: Tofacitinib: Double Blind Phase vs Placebo; General Health Subscale: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.4778, MMRM; LS mean difference = 1.77, 95% CI 2-sided [-3.18 to 6.72], Standard Error of Mean 2.48
Statistical Analysis 11: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Change in Health: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.8909, MMRM; LS mean difference = -0.02, 95% CI 2-sided [-0.28 to 0.25], Standard Error of Mean 0.13
Statistical Analysis 12: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Emotional Impact on Parent: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.1270, MMRM; LS mean difference = 8.97, 95% CI 2-sided [-2.61 to 20.55], Standard Error of Mean 5.81
Statistical Analysis 13: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Time Impact on Parent: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.0944, MMRM; LS mean difference = -6.72, 95% CI 2-sided [-14.62 to 1.18], Standard Error of Mean 3.96
Statistical Analysis 14: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Family Activities: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.0095, MMRM; LS mean difference = -8.60, 95% CI 2-sided [-15.03 to -2.17], Standard Error of Mean 3.23
Statistical Analysis 15: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Family Cohesion: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.5474, MMRM; LS mean difference = 2.59, 95% CI 2-sided [-5.96 to 11.14], Standard Error of Mean 4.29
Statistical Analysis 16: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Physical Health Summary: Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.0902, MMRM; LS mean difference = 3.48, 95% CI 2-sided [-0.56 to 7.52], Standard Error of Mean 2.03
Statistical Analysis 17: Comparison: Tofacitinib: Double Blind Phase vs Placebo; Psychosocial Health Summary : Analysis based on MMRM with fixed effects of treatment, visit, JIA category, open-label baseline CRP, treatment-by-visit interaction, and the Double-Blind baseline value; Test type: Superiority; p = 0.6539, MMRM; LS mean difference = -0.75, 95% CI 2-sided [-4.07 to 2.57], Standard Error of Mean 1.67

42. Secondary Outcome: Open Label Phase: Change From Baseline in Childhood Health Assessment Questionnaire (CHAQ)- Discomfort Index at Weeks 2, 4, 8, 12 and 18
Description: CHAQ is a validated instrument and comprises of two indices, Disability and Discomfort, and global assessment of arthritis (overall well-being). Discomfort Index included: assessment of discomfort, the parent/legal guardian/participant were asked to provide a response to the question: How much pain do you think your child had because of his or her illness in the past week?, The parent/legal guardian/ participant rated the overall pain on a 0 to 10 VAS, where '0' indicates 'No Pain' and '10' indicates 'Very Severe Pain', higher scores indicates more severity.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 184
score on scale
  Week 2: number analyzed (Participants) | 182
  Week 2 | -1.32 (2.10)
  Week 4: number analyzed (Participants) | 181
  Week 4 | -2.06 (2.16)
  Week 8: number analyzed (Participants) | 175
  Week 8 | -2.38 (2.40)
  Week 12: number analyzed (Participants) | 165
  Week 12 | -2.72 (2.28)
  Week 18: number analyzed (Participants) | 154
  Week 18 | -3.04 (2.57)

43. Secondary Outcome: Double Blind Phase:Change From Double-Blind Baseline in Childhood Health Assessment Questionnaire (CHAQ)- Discomfort Index at Weeks 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 42
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36,40 and 44
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 72 | 70
score on scale
  Week 20: number analyzed (Participants) | 71 | 70
  Week 20 | 0.08 (0.20) | 0.40 (0.20)
  Week 24: number analyzed (Participants) | 66 | 60
  Week 24 | -0.01 (0.24) | 0.94 (0.24)
  Week 28: number analyzed (Participants) | 63 | 49
  Week 28 | -0.23 (0.24) | 0.64 (0.25)
  Week 32: number analyzed (Participants) | 59 | 45
  Week 32 | 0.07 (0.27) | 1.06 (0.29)
  Week 36: number analyzed (Participants) | 55 | 37
  Week 36 | -0.21 (0.21) | 0.32 (0.24)
  Week 40: number analyzed (Participants) | 53 | 35
  Week 40 | -0.22 (0.24) | 0.49 (0.26)
  Week 44: number analyzed (Participants) | 49 | 33
  Week 44 | -0.36 (0.23) | 0.44 (0.25)
Statistical Analysis 1: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.1894, MMRM; LS Mean Difference = -0.32, 95% CI 2-sided [-0.80 to 0.16], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; p = 0.0026, MMRM; LS mean difference = -0.95, 95% CI 2-sided [-1.56 to -0.34], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; p = 0.0067, MMRM; LS mean difference = -0.87, 95% CI 2-sided [-1.50 to -0.25], Standard Error of Mean 0.31
Statistical Analysis 4: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority; p = 0.0091, MMRM; LS mean difference = -0.99, 95% CI 2-sided [-1.73 to -0.25], Standard Error of Mean 0.37
Statistical Analysis 5: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority; p = 0.0632, MMRM; LS mean difference = -0.53, 95% CI 2-sided [-1.09 to 0.03], Standard Error of Mean 0.28
Statistical Analysis 6: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority; p = 0.0306, MMRM; LS mean difference = -0.71, 95% CI 2-sided [-1.35 to -0.07], Standard Error of Mean 0.32
Statistical Analysis 7: Comparison: Tofacitinib: Double Blind Phase vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority; p = 0.0118, MMRM; LS mean difference = -0.80, 95% CI 2-sided [-1.41 to -0.18], Standard Error of Mean 0.31

44. Secondary Outcome: Open-Label Phase: Percentage of Participants With Active Uveitis at Baseline
Description: Uveitis is the inflammation of the uvea. Participants were assessed for presence of uveitis (according to Standard Uveitis Nomenclature [SUN]). If Uveitis was present in participant at Baseline, it was considered as "active uveitis"; If Uveitis was not present in participant at Baseline, it was considered as "Inactive uveitis". As per SUN, Uveitis is defined as: anterior (in which anterior chamber is primary site of inflammation); intermediate (primary site of inflammation: vitreous); posterior (primary site of inflammation: retina or choroid). Percentage of participants with active uveitis (of any type) are reported.
Time Frame: Baseline
Population: The OLFAS consists of all participants who were enrolled into open-label phase of the study and received at least one dose of study medication in open-label phase.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 225
percentage of participants | 0.0

45. Secondary Outcome: Double Blind Phase: Percentage of Participants With Active Uveitis at Week 24 and Week 44
Description: as for outcome 44
Time Frame: Week 24 and Week 44
Population: The double-blind safety analysis set (DBSAS) consists of all participants who have received at least one dose of study medication in double-blind phase.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 88 | 85
percentage of participants
  Week 24: Present | 0.0 | 1.2
  Week 44: Present | 0.0 | 0.0

46. Secondary Outcome: Open-Label Phase: Change From Baseline in the Tender Entheseal Assessment at Weeks 2, 4, 8, 12 and 18
Description: Participants with enthesitis-related arthritis (ERA) undergo Tender entheseal assessment. Tender entheseal assessment: Entheses were assessed and coded as: 1= any tenderness, 0= no tenderness, NE= not evaluable. Total number of tender entheses: 66*(total number of tender entheses with counts > 0)/number of non-missing tender entheses. If > 33 tender entheseal counts were missing, total number of tender entheses was defined as missing.
Time Frame: Baseline, weeks 2, 4, 8, 12 and 18
Population: OLERA included all participants who were enrolled into the open-label phase of study and received at least 1 dose of study medication in the open-label phase with ERA. Here, "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: tender entheses score
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 21
tender entheses score
  Week 2 | -1.57 (3.61)
  Week 4 | -2.52 (3.92)
  Week 8: number analyzed (Participants) | 20
  Week 8 | -3.05 (4.45)
  Week 12: number analyzed (Participants) | 20
  Week 12 | -3.15 (4.93)
  Week 18: number analyzed (Participants) | 20
  Week 18 | -3.50 (4.70)

47. Secondary Outcome: Double Blind Phase: Change From Double-Blind Baseline in the Tender Entheseal Assessment at Weeks 20, 24, 28, 32, 36, 40 and 44
Description: Participants with ERA undergo Tender entheseal assessment. Tender entheseal assessment: Entheses were assessed and coded as: 1= any tenderness, 0= no tenderness, NE= not evaluable. Total number of tender entheses: 66*(total number of tender entheses with counts > 0)/number of non-missing tender entheses. If > 33 tender entheseal counts were missing, total number of tender entheses was defined as missing.
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: DBERA included all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase with ERA. Here, "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: tender entheses score
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 9 | 7
tender entheses score
  Week 20 | 0.00 (0.87) | 0.86 (2.61)
  Week 24: number analyzed (Participants) | 9 | 5
  Week 24 | -1.00 (3.46) | 0.40 (2.19)
  Week 28: number analyzed (Participants) | 7 | 4
  Week 28 | -0.43 (2.57) | -0.75 (0.96)
  Week 32: number analyzed (Participants) | 6 | 4
  Week 32 | 0.33 (1.97) | 0.00 (0.82)
  Week 36: number analyzed (Participants) | 6 | 3
  Week 36 | -0.83 (2.04) | 0.33 (0.58)
  Week 40: number analyzed (Participants) | 5 | 3
  Week 40 | -2.00 (4.47) | 0.33 (0.58)
  Week 44: number analyzed (Participants) | 5 | 3
  Week 44 | -2.00 (5.66) | -0.33 (0.58)

48. Secondary Outcome: Open-Label Phase: Change From Baseline in the Modified Schober's Test at Week 2, 4, 8, 12 and 18
Description: Participants with ERA undergo Modified Schober's Test. In the Modified Schober's Test, a mark was placed 5 cm below the midpoint of a line that joined the posterior superior iliac spines. Another mark was placed 10 cm above the first. The participant then bent maximally forward with the knees fully extended. The distance between the two marks was then re-measured. The full measurement between the two lines was recorded to the nearest tenth of a centimeter and is reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 21
centimeter (cm)
  Week 2: number analyzed (Participants) | 16
  Week 2 | -0.35 (1.02)
  Week 4: number analyzed (Participants) | 15
  Week 4 | -0.20 (1.03)
  Week 8: number analyzed (Participants) | 16
  Week 8 | -0.12 (1.15)
  Week 12: number analyzed (Participants) | 16
  Week 12 | 0.02 (1.05)
  Week 18: number analyzed (Participants) | 16
  Week 18 | 0.29 (1.08)

49. Secondary Outcome: Double Blind Phase: Change From Double Blind Baseline in the Modified Schober's Test at Week 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 48
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 9 | 7
cm
  Week 20: number analyzed (Participants) | 7 | 5
  Week 20 | -0.46 (1.61) | -0.28 (0.47)
  Week 24: number analyzed (Participants) | 7 | 4
  Week 24 | -0.44 (1.27) | -0.35 (0.54)
  Week 28: number analyzed (Participants) | 5 | 3
  Week 28 | 0.32 (1.38) | -0.17 (0.57)
  Week 32: number analyzed (Participants) | 4 | 3
  Week 32 | 0.42 (1.84) | 0.63 (1.26)
  Week 36: number analyzed (Participants) | 3 | 2
  Week 36 | -0.53 (0.84) | 0.05 (0.21)
  Week 40: number analyzed (Participants) | 3 | 2
  Week 40 | 0.57 (1.62) | 0.85 (0.64)
  Week 44: number analyzed (Participants) | 3 | 2
  Week 44 | 0.50 (0.87) | 1.05 (2.47)

50. Secondary Outcome: Open-Label Phase: Change From Baseline in the Overall Back Pain and Nocturnal Back Pain Responses at Week 2, 4, 8, 12 and 18
Description: Participants with ERA undergo Overall Back Pain and Nocturnal Back Pain assessment. For Overall Back Pain, parent/legal guardian/participant were asked to provide a response to the question: What is the amount of back pain at any time that your child experienced in the past week? And For Nocturnal Back Pain: What is the amount of back pain at night that your child experienced in the past week?. Response to these questions was provided by parent/legal guardian/participant using a VAS of 0-10, where 0= No Pain and 10= Most Severe Pain, higher score indicated more severe pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 21
score on scale
  Week 2: Nocturnal Back Pain | -1.21 (3.10)
  Week 4: Nocturnal Back Pain | -1.33 (3.44)
  Week 8: Nocturnal Back Pain: number analyzed (Participants) | 20
  Week 8: Nocturnal Back Pain | -1.80 (3.18)
  Week 12: Nocturnal Back Pain: number analyzed (Participants) | 20
  Week 12: Nocturnal Back Pain | -2.30 (2.63)
  Week 18: Nocturnal Back Pain: number analyzed (Participants) | 20
  Week 18: Nocturnal Back Pain | -1.98 (2.94)
  Week 2: Overall back pain | -1.81 (2.89)
  Week 4: Overall back pain | -1.86 (3.29)
  Week 8:Overall back pain: number analyzed (Participants) | 20
  Week 8:Overall back pain | -2.65 (2.72)
  Week 12:Overall back pain: number analyzed (Participants) | 20
  Week 12:Overall back pain | -3.20 (2.54)
  Week 18: Overall back pain: number analyzed (Participants) | 20
  Week 18: Overall back pain | -3.30 (2.45)

51. Secondary Outcome: Double Blind Phase: Change From Double-Blind Baseline in the Overall Back Pain and Nocturnal Back Pain Responses at Week 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 50
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 9 | 7
score on scale
  Week 20: Nocturnal Back Pain | -0.17 (0.87) | 0.57 (0.93)
  Week 24: Nocturnal Back Pain: number analyzed (Participants) | 9 | 5
  Week 24: Nocturnal Back Pain | -1.06 (1.96) | 0.10 (0.42)
  Week 28: Nocturnal Back Pain: number analyzed (Participants) | 7 | 4
  Week 28: Nocturnal Back Pain | -0.79 (2.00) | 0.00 (0.41)
  Week 32: Nocturnal Back Pain: number analyzed (Participants) | 6 | 4
  Week 32: Nocturnal Back Pain | -1.58 (1.63) | 0.38 (0.63)
  Week 36: Nocturnal Back Pain: number analyzed (Participants) | 6 | 3
  Week 36: Nocturnal Back Pain | -0.75 (2.27) | 0.17 (0.29)
  Week 40: Nocturnal Back Pain: number analyzed (Participants) | 5 | 3
  Week 40: Nocturnal Back Pain | -2.00 (2.26) | 0.17 (0.29)
  Week 44: Nocturnal Back Pain: number analyzed (Participants) | 5 | 3
  Week 44: Nocturnal Back Pain | -0.80 (2.20) | 0.17 (0.29)
  Week 20: Overall back pain | 0.28 (1.89) | 0.57 (1.40)
  Week 24: Overall back pain: number analyzed (Participants) | 9 | 5
  Week 24: Overall back pain | 0.39 (2.10) | 0.00 (0.79)
  Week 28: Overall back pain: number analyzed (Participants) | 7 | 4
  Week 28: Overall back pain | 0.00 (2.60) | -0.25 (0.29)
  Week 32:Overall back pain: number analyzed (Participants) | 6 | 4
  Week 32:Overall back pain | -1.75 (2.25) | -0.13 (0.48)
  Week 36: Overall back pain: number analyzed (Participants) | 6 | 3
  Week 36: Overall back pain | 0.17 (1.29) | -0.50 (0.87)
  Week 40: Overall back pain: number analyzed (Participants) | 5 | 3
  Week 40: Overall back pain | 0.30 (1.79) | -0.50 (0.87)
  Week 44: Overall back pain: number analyzed (Participants) | 5 | 3
  Week 44: Overall back pain | -0.10 (3.45) | -0.50 (0.87)

52. Secondary Outcome: Open-Label Phase: Changes From Baseline in Percentage of Body Surface Area (BSA) Affected With Psoriasis at Weeks 2, 4, 8, 12 and 18
Description: Percentage of body surface area affected by psoriasis was estimated using the palm method. One of the participant's palm to proximal interphalangeal (PIP) and thumb =\together represented 1% of total BSA. Regions of the body were assigned specific number of palms with percentage (Head and Neck = 10% [10 palms], Upper extremities = 20% [20 palms], Trunk [axillae and groin] = 30% [30 palms], Lower extremities [buttocks] = 40% [40 palms]). The number of palms of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis. The total BSA affected was the summation of individual regions affected.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: OLPsA (OL psoriatic arthritis PsA) included all participants who were enrolled into the open-label phase of study and received at least 1 dose of study medication in the open-label phase with PsA. Here, "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 20
percentage of BSA
  Week 2 | 0.55 (4.70)
  Week 4: number analyzed (Participants) | 19
  Week 4 | -1.03 (2.49)
  Week 8: number analyzed (Participants) | 17
  Week 8 | -0.29 (6.11)
  Week 12: number analyzed (Participants) | 18
  Week 12 | -0.36 (5.93)
  Week 18: number analyzed (Participants) | 16
  Week 18 | -0.46 (6.48)

53. Secondary Outcome: Double Blind Phase: Changes From Double Blind Baseline in Body Surface Area (BSA) Affected With Psoriasis at Week 20, 24, 28, 32, 36, 40 and 44
Description: Percentage of body surface area affected by psoriasis was estimated using the palm method. One of the participant's palm to PIP and thumb together represented 1% of total BSA. Regions of the body were assigned specific number of palms with percentage (Head and Neck = 10% [10 palms], Upper extremities = 20% [20 palms], Trunk [axillae and groin] = 30% [30 palms], Lower extremities [buttocks] = 40% [40 palms]). The number of palms of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis. The total BSA affected was the summation of individual regions affected.
Time Frame: Double Blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: DBPsA included all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase with PsA. Here, "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 7 | 8
percentage of BSA
  Week 20: number analyzed (Participants) | 6 | 8
  Week 20 | -0.50 (1.22) | 0.28 (0.70)
  Week 24 | -0.14 (0.38) | 0.85 (1.71)
  Week 28: number analyzed (Participants) | 5 | 3
  Week 28 | -4.20 (8.84) | 0.33 (0.58)
  Week 32: number analyzed (Participants) | 5 | 3
  Week 32 | -0.60 (1.34) | 1.67 (2.89)
  Week 36: number analyzed (Participants) | 5 | 3
  Week 36 | -4.20 (8.90) | 1.33 (2.31)
  Week 40: number analyzed (Participants) | 5 | 3
  Week 40 | -4.60 (8.71) | 0.67 (1.15)
  Week 44: number analyzed (Participants) | 5 | 2
  Week 44 | -4.60 (8.71) | -0.05 (0.07)

54. Secondary Outcome: Open-Label Phase: Changes From Baseline in Physician's Global Assessment (PGA) of Psoriasis Assessments at Weeks 2, 4, 8, 12 and 18
Description: The PGA of psoriasis was scored on a 6-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 5 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and ranged as 0= no symptom to 5=severe, higher score indicates more severity.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: OLPsA included all participants who were enrolled into the open-label phase of study and received at least 1 dose of study medication in the open-label phase with PsA. Here, "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 20
score on scale
  Week 2 | -0.05 (0.39)
  Week 4: number analyzed (Participants) | 19
  Week 4 | -0.42 (0.84)
  Week 8: number analyzed (Participants) | 17
  Week 8 | -0.29 (0.92)
  Week 12: number analyzed (Participants) | 18
  Week 12 | -0.56 (0.86)
  Week 18: number analyzed (Participants) | 16
  Week 18 | -0.56 (1.03)

55. Secondary Outcome: Double Blind Phase:Change From Double-Blind Baseline in Physician's Global Assessment (PGA) of Psoriasis Assessments at Weeks 20, 24, 28, 32, 36, 40 and 44
Description: as for outcome 54
Time Frame: Double blind Baseline (Week 18), Weeks 20, 24, 28, 32, 36, 40 and 44
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 7 | 8
score on scale
  Week 20 | 0.14 (0.38) | 0.00 (0.00)
  Week 24 | 0.14 (0.38) | 0.38 (0.52)
  Week 28: number analyzed (Participants) | 5 | 3
  Week 28 | 0.20 (0.45) | 0.33 (0.58)
  Week 32: number analyzed (Participants) | 5 | 3
  Week 32 | 0.00 (0.00) | 0.33 (0.58)
  Week 36: number analyzed (Participants) | 5 | 3
  Week 36 | 0.00 (0.00) | 0.33 (0.58)
  Week 40: number analyzed (Participants) | 5 | 3
  Week 40 | 0.00 (0.00) | 0.00 (0.00)
  Week 44: number analyzed (Participants) | 5 | 2
  Week 44 | 0.00 (0.00) | -0.50 (0.71)

56. Secondary Outcome: Open-Label Phase: Taste Assessment of Tofacitinib Oral Solution on Day 14
Description: Oral solution was given only to participants weighing <40 kg and to the participants who were unable to swallow tablets. Taste assessment was evaluated using a 5 categories questionnaire. Participants were asked to answer in one of the following categories to describe the taste of oral solution of tofacitinib: dislike very much, dislike a little, not sure, like a little and like very much. Number of participants within each category are reported.
Time Frame: Day 14
Population: The OLFAS consists of all participants who were enrolled into open-label phase of the study and received at least one dose of study medication in open-label phase. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 84
Participants
  Dislike Very Much | 4
  Dislike a Little | 8
  Not Sure | 6
  Like a Little | 32
  Like Very Much | 34

57. Secondary Outcome: Open-Label Phase: Number of Participants With Serious Infections, Cytopenia, Malignancies and Cardiovascular Diseases
Description: Serious infection defined as any infection that requires hospitalization for treatment or requires parenteral antimicrobial therapy or meets other criteria that require it to be classified as a serious adverse event. Cytopenia was categorized as: lymphocyte counts: <500 lymphocytes/ millimeter^3 (mm), neutrophil counts <1000 neutrophils/mm^3, platelet counts <100,000 platelets/mm^3, any single hemoglobin value <8 grams/decilitre (g/dL) and any single hemoglobin value drops >=2 g/dL below baseline. Number of Participants With serious infections, cytopenia, malignancies and Cardiovascular Diseases are reported.
Time Frame: From the first dose of study drug up to Week 18
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 225
Participants
  Serious Infections | 3
  Cytopenia: Lymphocyte counts <500 lymphocytes/mm^3 | 1
  Cytopenia:Neutrophil counts <1000 neutrophils/mm^3 | 4
  Cytopenia: Platelet counts <100,000 platelets/mm^3 | 1
  Cytopenia: Any single hg value <8 g/dL | 1
  Cytopenia:Any hg value drops>=2g/dL below baseline | 17
  Malignancies | 0
  Cardiovascular Diseases | 0

58. Secondary Outcome: Double Blind Phase: Number of Participants With Serious Infections, Cytopenia, Malignancies and Cardiovascular Diseases
Description: Serious infection defined as any infection that requires hospitalization for treatment or requires parenteral antimicrobial therapy or meets other criteria that require it to be classified as a serious adverse event. Cytopenia was categorized as: lymphocyte counts <500 lymphocytes/mm^3, neutrophil counts <1000 neutrophils/mm^3, platelet counts <100000 platelets/mm^3, any single hemoglobin (hg) value <8 g/dL and any single hemoglobin value drops >=2 g/dL below baseline. Number of Participants With serious infections, cytopenia, malignancies and Cardiovascular Diseases are reported.
Time Frame: From the first dose of study drug in double blind up to week 44
Population: The DBFAS consists of all participants randomized to double-blind phase who received at least one dose of study medication in double-blind phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 88 | 85
Participants
  Serious Infections | 0 | 1
  Cytopenia: Lymphocyte counts <500 lymphocytes/mm^3 | 0 | 0
  Cytopenia:Neutrophil counts <1000 neutrophils/mm^3 | 0 | 2
  Cytopenia: Platelet counts <100,000 platelets/mm^3 | 1 | 0
  Cytopenia: Any single hemoglobin value <8 g/dL | 0 | 0
  Cytopenia: hg value drops >=2 g/dL below baseline | 3 | 7
  Malignancies | 0 | 0
  Cardiovascular Diseases | 0 | 0

59. Secondary Outcome: Open-Label Phase: Number of Participants With Tanner Staging Evaluation (Pubic Hair)
Description: Tanner stage is a scale used to document the stage of development of puberty by assessing the secondary sexual characteristics: Pubic hair (both male and female), breast size (for females); and size of the genitalia (for males).were assessed in this study and with values in the scale ranging from: Stage 1: no hair, Stage 2: downy hair, Stage 3: Scant terminal hair, Stage 4: Terminal hair that fills the entire triangle overlying the pubic region and Stage 5: Terminal hair that extends beyond the inguinal crease onto the thigh. Tanner Stage for pubic hair at Day 1 was summarized and reported using number of participants in each stage.
Time Frame: Day 1
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 218
Participants
  Stage 1 | 73
  Stage 2 | 21
  Stage 3 | 25
  Stage 4 | 47
  Stage 5 | 52

60. Secondary Outcome: Double Blind Phase: Number of Participants With Tanner Staging Evaluation (Pubic Hair)
Description: Tanner stage is a scale used to document the stage of development of puberty by assessing the secondary sexual characteristics: Pubic hair (both male and female), breast size (for females); and size of the genitalia (for males) were assessed in this study and with values in the scale ranging from: Stage 1: no hair, Stage 2: downy hair, Stage 3: Scant terminal hair, Stage 4: Terminal hair that fills the entire triangle overlying the pubic region and Stage 5: Terminal hair that extends beyond the inguinal crease onto the thigh. Tanner Stage for pubic hair at Week 44 was summarized and reported using number of participants in each stage.
Time Frame: Week 44
Population: The double-blind safety analysis set (DBSAS) consists of all participants who have received at least one dose of study medication in double-blind phase. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 56 | 38
Participants
  Stage 1 | 13 | 7
  Stage 2 | 8 | 7
  Stage 3 | 8 | 3
  Stage 4 | 14 | 4
  Stage 5 | 13 | 17

61. Secondary Outcome: Open-Label Phase: Number of Participants With Tanner Staging Evaluation (Breast Exam)
Description: Tanner stage is a scale used to document the stage of development of puberty by assessing the secondary sexual characteristics: Pubic hair (both male and female), breast size (for females); and size of the genitalia (for males).were assessed in this study and with values in the scale ranging from: Stage 1: No glandular breast tissue palpable, Stage 2: Breast bud palpable under areola (1st pubertal sign in females), Stage 3: Breast tissue palpable outside areola; no areolar development, Stage 4: Areola elevated above contour of the breast, forming "double scoop" appearance, Stage 5: Areolar mound recedes back into single breast contour with areolar hyperpigmentation, papillae development and nipple protrusion. Tanner Stage for Breast at Day 1 was summarized and reported using number of participants in each stage.
Time Frame: Day 1
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 163
Participants
  Stage 1 | 42
  Stage 2 | 19
  Stage 3 | 28
  Stage 4 | 34
  Stage 5 | 40

62. Secondary Outcome: Double Blind Phase: Number of Participants With Tanner Staging Evaluation (Breast Exam)
Description: Tanner stage is a scale used to document the stage of development of puberty by assessing the secondary sexual characteristics: Pubic hair (both male and female), breast size (for females); and size of the genitalia (for males).were assessed in this study and with values in the scale ranging from: Stage 1: No glandular breast tissue palpable, Stage 2: Breast bud palpable under areola (1st pubertal sign in females), Stage 3: Breast tissue palpable outside areola; no areolar development, Stage 4: Areola elevated above contour of the breast, forming "double scoop" appearance, Stage 5: Areolar mound recedes back into single breast contour with areolar hyperpigmentation, papillae development and nipple protrusion. Tanner Stage for Breast at Week 44 was summarized and reported using number of participants in each stage.
Time Frame: Week 44
Population: The DBSAS consists of all participants who have received at least one dose of study medication in double-blind phase. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 43 | 28
Participants
  Stage 1 | 6 | 8
  Stage 2 | 8 | 2
  Stage 3 | 7 | 2
  Stage 4 | 13 | 3
  Stage 5 | 9 | 13

63. Secondary Outcome: Open-Label Phase: Number of Participants With Tanner Staging Evaluation (Genitalia)
Description: Tanner stage is a scale used to document the stage of development of puberty by assessing the secondary sexual characteristics: Pubic hair (both male and female), breast size (for females); and size of the genitalia (for males).were assessed in this study and with values in the scale ranging from: Stage 1: Testicular volume < 4 ml or long axis < 2.5 cm, Stage 2: 4 ml-8 ml (or 2.5-3.3 cm long), 1st pubertal sign in males, Stage 3: 9 ml-12 ml (or 3.4-4.0 cm long), Stage 4: 15-20 ml (or 4.1-4.5 cm long), Stage 5: > 20 ml (or > 4.5 cm long). Tanner Stage for genitalia at Day 1 was summarized and reported using number of participants in each stage.
Time Frame: Day 1
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 55
Participants
  Stage 1 | 24
  Stage 2 | 6
  Stage 3 | 8
  Stage 4 | 11
  Stage 5 | 6

64. Secondary Outcome: Double Blind Phase: Number of Participants With Tanner Staging Evaluation (Genitalia)
Description: Tanner stage is a scale used to document the stage of development of puberty by assessing the secondary sexual characteristics: Pubic hair (both male and female), breast size (for females); and size of the genitalia (for males).were assessed in this study and with values in the scale ranging from: Stage 1: Testicular volume < 4 ml or long axis < 2.5 cm, Stage 2: 4 ml-8 ml (or 2.5-3.3 cm long), 1st pubertal sign in males, Stage 3: 9 ml-12 ml (or 3.4-4.0 cm long), Stage 4: 15-20 ml (or 4.1-4.5 cm long), Stage 5: > 20 ml (or > 4.5 cm long). Tanner Stage for genitalia at Week 44 was summarized and reported using number of participants in each stage.
Time Frame: Week 44
Population: The DBSAS consists of all participants who have received atleast one dose of study medication in double-blind phase. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 13 | 10
Participants
  Stage 1 | 5 | 0
  Stage 2 | 0 | 5
  Stage 3 | 2 | 0
  Stage 4 | 5 | 1
  Stage 5 | 1 | 4

65. Secondary Outcome: Open-Label Phase: Number of Participants With Laboratory Abnormalities
Description: Criteria: Hemoglobin(Hg),hematocrit erythrocytes(Ery); <0.8*lower limit of normal (LLN), Ery. Mean Corpuscular Volume; <0.9*LLN, >1.1*upper limit of normal (ULN), Platelets; <0.5*LLN, >1.75*ULN, Leukocytes (leu); <0.6*LLN, >1.5*ULN, Lymphocytes (Ly), Ly/leu, Neutrophils, Neutrophils/leu <0.8*LLN, Basophils/leu, Eosinophils, Eosinophils/leu, Monocytes, Monocytes/leu >1.2*ULN, Ery Sedimentation Rate >1.5*ULN. Bilirubin, Indirect Bilirubin >1.5*ULN, AST, ALT, Gamma Glutamyl Transferase, Alkaline Phosphatase >3.0*ULN, Albumin >1.2*ULN, Creatinine >1.3*ULN, HDL Cholesterol (Chol)<0.8*LLN, LDL Chol, LDL Chol Friedewald Est PEG >1.2*ULN, Triglycerides >1.3*ULN, Calcium <0.9*LLN, Bicarbonate <0.9*LLN, Glucose >1.5*ULN, Creatine Kinase >2.0*ULN, C Reactive Protein >1.1*ULN, Chol >1.3*ULN. Urinalysis: Specific Gravity >1.030, Glucose, Ketones, Protein, Hg, Nitrite, Leu Esterase >=1, Ery, Leu >=20, Hyaline Casts >1.Only those category in which at least 1 participant had data is reported.
Time Frame: From the first dose of study drug up to Week 18
Population: The OLFAS consists of all participants who were enrolled into open-label phase of the study and received at least one dose of study medication in open-label phase. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 225
Participants
  Hemoglobin (<0.8* LLN): number analyzed (Participants) | 224
  Hemoglobin (<0.8* LLN) | 1
  Hematocrit (<0.8* LLN): number analyzed (Participants) | 224
  Hematocrit (<0.8* LLN) | 1
  Erythrocytes (<0.8* LLN): number analyzed (Participants) | 224
  Erythrocytes (<0.8* LLN) | 2
  Ery. Mean Corpuscular Volume (<0.9*LLN): number analyzed (Participants) | 224
  Ery. Mean Corpuscular Volume (<0.9*LLN) | 3
  Ery. Mean Corpuscular Volume (>1.1*ULN ): number analyzed (Participants) | 224
  Ery. Mean Corpuscular Volume (>1.1*ULN ) | 4
  Platelets (<0.5*LLN): number analyzed (Participants) | 224
  Platelets (<0.5*LLN) | 1
  Platelets (>1.75*ULN): number analyzed (Participants) | 224
  Platelets (>1.75*ULN) | 2
  Leukocytes (<0.6*LLN): number analyzed (Participants) | 224
  Leukocytes (<0.6*LLN) | 1
  Leukocytes (>1.5*ULN): number analyzed (Participants) | 224
  Leukocytes (>1.5*ULN) | 2
  Lymphocytes (<0.8*LLN): number analyzed (Participants) | 224
  Lymphocytes (<0.8*LLN) | 7
  Lymphocytes (>1.2*ULN): number analyzed (Participants) | 224
  Lymphocytes (>1.2*ULN) | 2
  Lymphocytes/Leukocytes (<0.8*LLN): number analyzed (Participants) | 224
  Lymphocytes/Leukocytes (<0.8*LLN) | 15
  Lymphocytes/Leukocytes (>1.2*ULN): number analyzed (Participants) | 224
  Lymphocytes/Leukocytes (>1.2*ULN) | 20
  Neutrophils (<0.8*LLN): number analyzed (Participants) | 224
  Neutrophils (<0.8*LLN) | 8
  Neutrophils (>1.2*ULN): number analyzed (Participants) | 224
  Neutrophils (>1.2*ULN) | 18
  Neutrophils/Leukocytes (<0.8*LLN): number analyzed (Participants) | 224
  Neutrophils/Leukocytes (<0.8*LLN) | 19
  Basophils/Leukocytes (>1.2*ULN): number analyzed (Participants) | 224
  Basophils/Leukocytes (>1.2*ULN) | 37
  Eosinophils (>1.2*ULN): number analyzed (Participants) | 224
  Eosinophils (>1.2*ULN) | 53
  Eosinophils/Leukocytes (>1.2*ULN): number analyzed (Participants) | 224
  Eosinophils/Leukocytes (>1.2*ULN) | 32
  Monocytes (>1.2*ULN): number analyzed (Participants) | 224
  Monocytes (>1.2*ULN) | 3
  Monocytes/Leukocytes (>1.2*ULN): number analyzed (Participants) | 224
  Monocytes/Leukocytes (>1.2*ULN) | 38
  Ery. Sedimentation Rate (>1.5*ULN): number analyzed (Participants) | 224
  Ery. Sedimentation Rate (>1.5*ULN) | 65
  Bilirubin (>1.5*ULN) | 1
  Indirect Bilirubin (>1.5*ULN) | 1
  Aspartate Aminotransferase (AST) (>3.0*ULN) | 4
  Alanine Aminotransferase (ALT) (>3.0*ULN) | 5
  GGT (>3.0*ULN) | 1
  Alkaline Phosphatase (>3.0*ULN) | 1
  Albumin (>1.2*ULN) | 1
  Creatinine (>1.3*ULN) | 1
  HDL Cholesterol (<0.8*LLN): number analyzed (Participants) | 223
  HDL Cholesterol (<0.8*LLN) | 2
  LDL Cholesterol (>1.2*ULN): number analyzed (Participants) | 87
  LDL Cholesterol (>1.2*ULN) | 4
  LDL Chol Friedewald Est PEG (>1.2*ULN): number analyzed (Participants) | 222
  LDL Chol Friedewald Est PEG (>1.2*ULN) | 1
  Triglycerides (>1.3*ULN): number analyzed (Participants) | 222
  Triglycerides (>1.3*ULN) | 27
  Calcium (<0.9*LLN) | 1
  Bicarbonate (<0.9*LLN) | 10
  Glucose (>1.5*ULN) | 2
  Creatine Kinase (>2.0*ULN): number analyzed (Participants) | 224
  Creatine Kinase (>2.0*ULN) | 12
  C Reactive Protein (>1.1*ULN) | 122
  Cholesterol (>1.3*ULN): number analyzed (Participants) | 223
  Cholesterol (>1.3*ULN) | 2
  Specific Gravity (>1.030) | 32
  URINE Glucose (>=1) | 1
  Ketones (>=1) | 11
  URINE Protein (>=1) | 9
  URINE Hemoglobin (>=1) | 48
  Nitrite (>=1) | 6
  Leukocyte Esterase (>=1) | 59
  URINE Erythrocytes (>=1): number analyzed (Participants) | 113
  URINE Erythrocytes (>=1) | 23
  URINE Leukocytes (>=20): number analyzed (Participants) | 150
  URINE Leukocytes (>=20) | 16
  Hyaline Casts (>1): number analyzed (Participants) | 3
  Hyaline Casts (>1) | 1

66. Secondary Outcome: Double Blind Phase: Number of Participants With Laboratory Abnormalities
Description: Criteria: Hg, hematocrit Ery; <0.8* LLN, Ery. Mean Corpuscular Volume; <0.9*LLN, >1.1* ULN, Platelets; <0.5*LLN, >1.75*ULN, leu; <0.6*LLN, >1.5*ULN, Ly, Ly/leu, Neutrophils, Neutrophils/leu <0.8*LLN, Basophils/leu, Eosinophils, Eosinophils/leu, Monocytes, Monocytes/leu >1.2*ULN, Prothrombin Time >1.1*ULN, Ery Sedimentation Rate >1.5*ULN. Bilirubin, Direct Bilirubin, Indirect Bilirubin >1.5*ULN, AST, ALT, Gamma Glutamyl Transferase (GGT), Alkaline Phosphatase >3.0*ULN, Albumin >1.2*ULN, Creatinine >1.3*ULN, HDL Cholesterol (Chol)<0.8*LLN, LDL Chol, LDL Chol Friedewald Est PEG >1.2*ULN, Triglycerides >1.3*ULN, Calcium <0.9*LLN, Bicarbonate <0.9*LLN, Glucose >1.5*ULN, Creatine Kinase >2.0*ULN, C Reactive Protein >1.1*ULN, Chol >1.3*ULN. Urinalysis: Specific Gravity >1.030, pH >8, urine Glucose, Ketones, Protein, Hg, Nitrite, Leu Esterase >=1, Ery, Leu >=20, Hyaline Casts >1.Only those category in which at least 1 participant had data is reported.
Time Frame: From the first dose of study drug in double blind up to Week 44
Population: The DBSAS consists of all participants who have received atleast one dose of study medication in double-blind phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 88 | 85
Participants
  Hemoglobin (<0.8*LLN): number analyzed (Participants) | 87 | 85
  Hemoglobin (<0.8*LLN) | 1 | 3
  Hematocrit (<0.8*LLN): number analyzed (Participants) | 87 | 85
  Hematocrit (<0.8*LLN) | 0 | 2
  Erythrocytes (<0.8*LLN): number analyzed (Participants) | 87 | 85
  Erythrocytes (<0.8*LLN) | 0 | 2
  Ery. Mean Corpuscular Volume (<0.9*LLN): number analyzed (Participants) | 87 | 85
  Ery. Mean Corpuscular Volume (<0.9*LLN) | 2 | 1
  Ery. Mean Corpuscular Volume (>1.1*ULN): number analyzed (Participants) | 87 | 85
  Ery. Mean Corpuscular Volume (>1.1*ULN) | 1 | 2
  Platelets (<0.5*LLN): number analyzed (Participants) | 88 | 84
  Platelets (<0.5*LLN) | 1 | 0
  Leukocytes (<0.6*LLN): number analyzed (Participants) | 87 | 85
  Leukocytes (<0.6*LLN) | 0 | 1
  Leukocytes (>1.5*ULN): number analyzed (Participants) | 87 | 85
  Leukocytes (>1.5*ULN) | 1 | 0
  Lymphocytes (<0.8*LLN): number analyzed (Participants) | 87 | 85
  Lymphocytes (<0.8*LLN) | 5 | 1
  Lymphocytes (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Lymphocytes (>1.2*ULN) | 1 | 0
  Lymphocytes/Leukocytes (<0.8*LLN): number analyzed (Participants) | 87 | 85
  Lymphocytes/Leukocytes (<0.8*LLN) | 9 | 5
  Lymphocytes/Leukocytes (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Lymphocytes/Leukocytes (>1.2*ULN) | 5 | 7
  Neutrophils (<0.8*LLN): number analyzed (Participants) | 87 | 85
  Neutrophils (<0.8*LLN) | 1 | 3
  Neutrophils (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Neutrophils (>1.2*ULN) | 7 | 5
  Neutrophils/Leukocytes (<0.8*LLN): number analyzed (Participants) | 87 | 85
  Neutrophils/Leukocytes (<0.8*LLN) | 5 | 6
  Basophils (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Basophils (>1.2*ULN) | 1 | 0
  Basophils/Leukocytes (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Basophils/Leukocytes (>1.2*ULN) | 14 | 15
  Eosinophils (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Eosinophils (>1.2*ULN) | 27 | 18
  Eosinophils/Leukocytes (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Eosinophils/Leukocytes (>1.2*ULN) | 21 | 14
  Monocytes (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Monocytes (>1.2*ULN) | 2 | 2
  Monocytes/Leukocytes (>1.2*ULN): number analyzed (Participants) | 87 | 85
  Monocytes/Leukocytes (>1.2*ULN) | 18 | 19
  Prothrombin Time (>1.1*ULN): number analyzed (Participants) | 3 | 2
  Prothrombin Time (>1.1*ULN) | 0 | 1
  Ery. Sedimentation Rate (>1.5*ULN) | 26 | 19
  Bilirubin (>1.5*ULN) | 1 | 0
  Direct Bilirubin (>1.5*ULN) | 1 | 0
  Indirect Bilirubin (>1.5*ULN) | 1 | 0
  Alanine Aminotransferase(>3.0*ULN) | 1 | 2
  GGT (>3.0*ULN) | 1 | 0
  HDL Cholesterol (<0.8*LLN): number analyzed (Participants) | 70 | 61
  HDL Cholesterol (<0.8*LLN) | 0 | 2
  Triglycerides (>1.3*ULN): number analyzed (Participants) | 71 | 61
  Triglycerides (>1.3*ULN) | 8 | 6
  Potassium (>1.1*ULN) | 1 | 0
  Calcium (<0.9*LLN ) | 1 | 1
  Glucose (>1.5*ULN) | 1 | 0
  Creatine Kinase (>2.0*ULN) | 2 | 2
  C Reactive Protein (>1.1*ULN) | 44 | 47
  Specific Gravity (>1.030) | 12 | 7
  pH (>8) | 0 | 1
  URINE Glucose (>=1) | 1 | 1
  Ketones (>=1) | 7 | 10
  URINE Protein (>=1) | 4 | 4
  URINE Hemoglobin (>=1) | 25 | 11
  Nitrite (>=1) | 3 | 6
  Leukocyte Esterase (>=1) | 26 | 25
  URINE Erythrocytes (>=20): number analyzed (Participants) | 51 | 41
  URINE Erythrocytes (>=20) | 10 | 6
  URINE Leukocytes (>=20): number analyzed (Participants) | 66 | 57
  URINE Leukocytes (>=20) | 6 | 6
  Hyaline Casts (>1): number analyzed (Participants) | 2 | 1
  Hyaline Casts (>1) | 1 | 1
  Granular Casts (>1): number analyzed (Participants) | 0 | 1
  Granular Casts (>1) | 0 | 1
  Bicarbonate (<0.9*LLN) | 0 | 2

67. Secondary Outcome: Open-Label Phase: Number of Participants With Physical Examination Abnormalities
Description: Physical examination included: abdomen, ears, extremities, eyes, general appearance, head, heart, lungs, lymph nodes, neurological, nose, skin, and throat. Abnormality in physical examination was based on investigator's discretion.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 18
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 225
Participants
  Abdomen: Baseline | 1
  Abdomen: Week 2: number analyzed (Participants) | 223
  Abdomen: Week 2 | 2
  Abdomen: Week 4: number analyzed (Participants) | 218
  Abdomen: Week 4 | 3
  Abdomen: Week 8: number analyzed (Participants) | 214
  Abdomen: Week 8 | 2
  Abdomen: Week 12: number analyzed (Participants) | 203
  Abdomen: Week 12 | 2
  Abdomen: Week 18: number analyzed (Participants) | 189
  Abdomen: Week 18 | 1
  Ears: Baseline | 5
  Ears: Week 2: number analyzed (Participants) | 1
  Ears: Week 2 | 0
  Ears: Week 4: number analyzed (Participants) | 2
  Ears: Week 4 | 0
  Ears: Week 8: number analyzed (Participants) | 9
  Ears: Week 8 | 0
  Ears: Week 12: number analyzed (Participants) | 10
  Ears: Week 12 | 0
  Ears: Week 18: number analyzed (Participants) | 189
  Ears: Week 18 | 3
  Extremities: Baseline | 49
  Extremities: Week 2: number analyzed (Participants) | 223
  Extremities: Week 2 | 43
  Extremities: Week 4: number analyzed (Participants) | 218
  Extremities: Week 4 | 35
  Extremities: Week 8: number analyzed (Participants) | 214
  Extremities: Week 8 | 30
  Extremities: Week 12: number analyzed (Participants) | 203
  Extremities: Week 12 | 28
  Extremities: Week 18: number analyzed (Participants) | 189
  Extremities: Week 18 | 23
  Eyes: Baseline | 2
  Eyes: Week 2: number analyzed (Participants) | 1
  Eyes: Week 2 | 0
  Eyes: Week 4: number analyzed (Participants) | 2
  Eyes: Week 4 | 0
  Eyes: Week 8: number analyzed (Participants) | 9
  Eyes: Week 8 | 0
  Eyes: Week 12: number analyzed (Participants) | 10
  Eyes: Week 12 | 0
  Eyes: Week 18: number analyzed (Participants) | 189
  Eyes: Week 18 | 2
  General appearance: Baseline | 16
  General appearance: Week 2: number analyzed (Participants) | 1
  General appearance: Week 2 | 0
  General appearance: Week 4: number analyzed (Participants) | 2
  General appearance: Week 4 | 1
  General appearance: Week 8: number analyzed (Participants) | 9
  General appearance: Week 8 | 2
  General appearance: Week 12: number analyzed (Participants) | 10
  General appearance: Week 12 | 0
  General appearance: Week 18: number analyzed (Participants) | 189
  General appearance: Week 18 | 5
  Head: Baseline | 3
  Head: Week 2: number analyzed (Participants) | 1
  Head: Week 2 | 0
  Head: Week 4: number analyzed (Participants) | 2
  Head: Week 4 | 0
  Head: Week 8: number analyzed (Participants) | 9
  Head: Week 8 | 0
  Head: Week 12: number analyzed (Participants) | 10
  Head: Week 12 | 0
  Head: Week 18: number analyzed (Participants) | 189
  Head: Week 18 | 4
  Heart: Baseline | 0
  Heart: Week 2: number analyzed (Participants) | 223
  Heart: Week 2 | 0
  Heart: Week 4: number analyzed (Participants) | 218
  Heart: Week 4 | 0
  Heart: Week 8: number analyzed (Participants) | 214
  Heart: Week 8 | 2
  Heart: Week 12: number analyzed (Participants) | 203
  Heart: Week 12 | 0
  Heart: Week 18: number analyzed (Participants) | 189
  Heart: Week 18 | 0
  Lungs: Baseline | 1
  Lungs: Week 2: number analyzed (Participants) | 223
  Lungs: Week 2 | 1
  Lungs: Week 4: number analyzed (Participants) | 218
  Lungs: Week 4 | 0
  Lungs: Week 8: number analyzed (Participants) | 214
  Lungs: Week 8 | 1
  Lungs: Week 12: number analyzed (Participants) | 203
  Lungs: Week 12 | 1
  Lungs: Week 18: number analyzed (Participants) | 189
  Lungs: Week 18 | 0
  Lymph nodes: Baseline | 2
  Lymph nodes: Week 2: number analyzed (Participants) | 223
  Lymph nodes: Week 2 | 5
  Lymph nodes: Week 4: number analyzed (Participants) | 218
  Lymph nodes: Week 4 | 5
  Lymph nodes: Week 8: number analyzed (Participants) | 214
  Lymph nodes: Week 8 | 5
  Lymph nodes: Week 12: number analyzed (Participants) | 203
  Lymph nodes: Week 12 | 3
  Lymph nodes: Week 18: number analyzed (Participants) | 189
  Lymph nodes: Week 18 | 4
  Neurological: Baseline | 4
  Neurological: Week 2: number analyzed (Participants) | 1
  Neurological: Week 2 | 1
  Neurological: Week 4: number analyzed (Participants) | 2
  Neurological: Week 4 | 0
  Neurological: Week 8: number analyzed (Participants) | 9
  Neurological: Week 8 | 0
  Neurological: Week 12: number analyzed (Participants) | 10
  Neurological: Week 12 | 0
  Neurological: Week 18: number analyzed (Participants) | 189
  Neurological: Week 18 | 4
  Nose: Baseline | 0
  Nose: Week 2: number analyzed (Participants) | 1
  Nose: Week 2 | 0
  Nose: Week 4: number analyzed (Participants) | 2
  Nose: Week 4 | 0
  Nose: Week 8: number analyzed (Participants) | 9
  Nose: Week 8 | 0
  Nose: Week 12: number analyzed (Participants) | 10
  Nose: Week 12 | 0
  Nose: Week 18: number analyzed (Participants) | 189
  Nose: Week 18 | 5
  Skin: Baseline | 27
  Skin: Week 2: number analyzed (Participants) | 1
  Skin: Week 2 | 0
  Skin: Week 4: number analyzed (Participants) | 2
  Skin: Week 4 | 1
  Skin: Week 8: number analyzed (Participants) | 9
  Skin: Week 8 | 1
  Skin: Week 12: number analyzed (Participants) | 10
  Skin: Week 12 | 0
  Skin: Week 18: number analyzed (Participants) | 189
  Skin: Week 18 | 12
  Throat: Baseline | 1
  Throat: Week 2: number analyzed (Participants) | 1
  Throat: Week 2 | 0
  Throat: Week 4: number analyzed (Participants) | 2
  Throat: Week 4 | 0
  Throat: Week 8: number analyzed (Participants) | 9
  Throat: Week 8 | 0
  Throat: Week 12: number analyzed (Participants) | 10
  Throat: Week 12 | 0
  Throat: Week 18: number analyzed (Participants) | 189
  Throat: Week 18 | 6

68. Secondary Outcome: Double Blind Phase: Number of Participants With Physical Examination Abnormalities
Description: as for outcome 67
Time Frame: Weeks 18, 20, 24, 28, 32, 36, 40 and 44
Population: The DBSAS consists of all participants who have received at least one dose of study medication in double-blind phase. Here, 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 88 | 85
Participants
  Abdomen: Week 18: number analyzed (Participants) | 88 | 84
  Abdomen: Week 18 | 0 | 1
  Abdomen: Week 20: number analyzed (Participants) | 87 | 85
  Abdomen: Week 20 | 1 | 1
  Abdomen: Week 24: number analyzed (Participants) | 82 | 73
  Abdomen: Week 24 | 1 | 1
  Abdomen: Week 28: number analyzed (Participants) | 75 | 57
  Abdomen: Week 28 | 0 | 0
  Abdomen: Week 32: number analyzed (Participants) | 70 | 52
  Abdomen: Week 32 | 0 | 0
  Abdomen: Week 36: number analyzed (Participants) | 66 | 43
  Abdomen: Week 36 | 0 | 0
  Abdomen: Week 40: number analyzed (Participants) | 63 | 41
  Abdomen: Week 40 | 0 | 0
  Abdomen: Week 44: number analyzed (Participants) | 59 | 38
  Abdomen: Week 44 | 0 | 0
  Ears: Week 18: number analyzed (Participants) | 88 | 84
  Ears: Week 18 | 3 | 0
  Ears: Week 20: number analyzed (Participants) | 4 | 5
  Ears: Week 20 | 0 | 0
  Ears: Week 24: number analyzed (Participants) | 5 | 5
  Ears: Week 24 | 0 | 0
  Ears: Week 28: number analyzed (Participants) | 2 | 2
  Ears: Week 28 | 0 | 0
  Ears: Week 32: number analyzed (Participants) | 2 | 3
  Ears: Week 32 | 0 | 0
  Ears: Week 40: number analyzed (Participants) | 1 | 1
  Ears: Week 40 | 0 | 1
  Ears: Week 44: number analyzed (Participants) | 59 | 38
  Ears: Week 44 | 0 | 0
  Extremities: Week 18: number analyzed (Participants) | 88 | 84
  Extremities: Week 18 | 9 | 12
  Extremities: Week 20: number analyzed (Participants) | 87 | 85
  Extremities: Week 20 | 11 | 14
  Extremities: Week 24: number analyzed (Participants) | 82 | 73
  Extremities: Week 24 | 5 | 7
  Extremities: Week 28: number analyzed (Participants) | 75 | 57
  Extremities: Week 28 | 6 | 6
  Extremities: Week 32: number analyzed (Participants) | 70 | 52
  Extremities: Week 32 | 1 | 8
  Extremities: Week 36: number analyzed (Participants) | 66 | 43
  Extremities: Week 36 | 2 | 6
  Extremities: Week 40: number analyzed (Participants) | 63 | 41
  Extremities: Week 40 | 3 | 6
  Extremities: Week 44: number analyzed (Participants) | 59 | 38
  Extremities: Week 44 | 3 | 7
  Eyes: Week 18: number analyzed (Participants) | 88 | 84
  Eyes: Week 18 | 2 | 0
  Eyes: Week 20: number analyzed (Participants) | 4 | 5
  Eyes: Week 20 | 0 | 0
  Eyes: Week 24: number analyzed (Participants) | 5 | 5
  Eyes: Week 24 | 0 | 0
  Eyes: Week 28: number analyzed (Participants) | 2 | 2
  Eyes: Week 28 | 0 | 0
  Eyes: Week 32: number analyzed (Participants) | 2 | 3
  Eyes: Week 32 | 0 | 0
  Eyes: Week 40: number analyzed (Participants) | 1 | 1
  Eyes: Week 40 | 0 | 0
  Eyes: Week 44: number analyzed (Participants) | 59 | 38
  Eyes: Week 44 | 1 | 0
  General appearance: Week 18: number analyzed (Participants) | 88 | 84
  General appearance: Week 18 | 2 | 3
  General appearance: Week 20: number analyzed (Participants) | 4 | 5
  General appearance: Week 20 | 1 | 1
  General appearance: Week 24: number analyzed (Participants) | 5 | 5
  General appearance: Week 24 | 0 | 0
  General appearance: Week 28: number analyzed (Participants) | 2 | 2
  General appearance: Week 28 | 0 | 0
  General appearance: Week 32: number analyzed (Participants) | 2 | 3
  General appearance: Week 32 | 0 | 0
  General appearance: Week 40: number analyzed (Participants) | 1 | 1
  General appearance: Week 40 | 0 | 0
  General appearance: Week 44: number analyzed (Participants) | 59 | 38
  General appearance: Week 44 | 1 | 0
  Head: Week 18: number analyzed (Participants) | 88 | 84
  Head: Week 18 | 3 | 1
  Head: Week 20: number analyzed (Participants) | 4 | 5
  Head: Week 20 | 0 | 0
  Head: Week 24: number analyzed (Participants) | 5 | 5
  Head: Week 24 | 0 | 0
  Head: Week 28: number analyzed (Participants) | 2 | 2
  Head: Week 28 | 0 | 0
  Head: Week 32: number analyzed (Participants) | 2 | 3
  Head: Week 32 | 0 | 1
  Head: Week 40: number analyzed (Participants) | 1 | 1
  Head: Week 40 | 1 | 0
  Head: Week 44: number analyzed (Participants) | 59 | 38
  Head: Week 44 | 0 | 0
  Heart: Week 18: number analyzed (Participants) | 88 | 84
  Heart: Week 18 | 0 | 0
  Heart: Week 20: number analyzed (Participants) | 87 | 85
  Heart: Week 20 | 0 | 0
  Heart: Week 24: number analyzed (Participants) | 82 | 73
  Heart: Week 24 | 0 | 0
  Heart: Week 28: number analyzed (Participants) | 75 | 57
  Heart: Week 28 | 0 | 0
  Heart: Week 32: number analyzed (Participants) | 70 | 52
  Heart: Week 32 | 0 | 0
  Heart: Week 36: number analyzed (Participants) | 66 | 43
  Heart: Week 36 | 0 | 0
  Heart: Week 40: number analyzed (Participants) | 63 | 41
  Heart: Week 40 | 0 | 0
  Heart: Week 44: number analyzed (Participants) | 59 | 38
  Heart: Week 44 | 0 | 0
  Lungs: Week 18: number analyzed (Participants) | 88 | 84
  Lungs: Week 18 | 0 | 0
  Lungs: Week 20: number analyzed (Participants) | 87 | 85
  Lungs: Week 20 | 1 | 0
  Lungs: Week 24: number analyzed (Participants) | 82 | 73
  Lungs: Week 24 | 1 | 0
  Lungs: Week 28: number analyzed (Participants) | 75 | 57
  Lungs: Week 28 | 1 | 0
  Lungs: Week 32: number analyzed (Participants) | 70 | 52
  Lungs: Week 32 | 0 | 0
  Lungs: Week 36: number analyzed (Participants) | 66 | 43
  Lungs: Week 36 | 0 | 0
  Lungs: Week 40: number analyzed (Participants) | 63 | 41
  Lungs: Week 40 | 0 | 1
  Lungs: Week 44: number analyzed (Participants) | 59 | 38
  Lungs: Week 44 | 0 | 0
  Lymph nodes: Week 18: number analyzed (Participants) | 88 | 84
  Lymph nodes: Week 18 | 3 | 1
  Lymph nodes: Week 20: number analyzed (Participants) | 87 | 85
  Lymph nodes: Week 20 | 3 | 0
  Lymph nodes: Week 24: number analyzed (Participants) | 82 | 73
  Lymph nodes: Week 24 | 2 | 1
  Lymph nodes: Week 28: number analyzed (Participants) | 75 | 57
  Lymph nodes: Week 28 | 1 | 0
  Lymph nodes: Week 32: number analyzed (Participants) | 70 | 52
  Lymph nodes: Week 32 | 1 | 1
  Lymph nodes: Week 36: number analyzed (Participants) | 66 | 43
  Lymph nodes: Week 36 | 1 | 0
  Lymph nodes: Week 40: number analyzed (Participants) | 63 | 41
  Lymph nodes: Week 40 | 2 | 0
  Lymph nodes: Week 44: number analyzed (Participants) | 59 | 38
  Lymph nodes: Week 44 | 1 | 1
  Neurological: Week 18 | 3 | 1
  Neurological: Week 20: number analyzed (Participants) | 4 | 5
  Neurological: Week 20 | 1 | 0
  Neurological: Week 24: number analyzed (Participants) | 5 | 5
  Neurological: Week 24 | 0 | 0
  Neurological: Week 28: number analyzed (Participants) | 2 | 2
  Neurological: Week 28 | 0 | 0
  Neurological: Week 32: number analyzed (Participants) | 2 | 3
  Neurological: Week 32 | 0 | 0
  Neurological: Week 40: number analyzed (Participants) | 1 | 1
  Neurological: Week 40 | 0 | 0
  Neurological: Week 44: number analyzed (Participants) | 59 | 38
  Neurological: Week 44 | 1 | 1
  Nose: Week 18: number analyzed (Participants) | 88 | 84
  Nose: Week 18 | 4 | 0
  Nose: Week 20: number analyzed (Participants) | 4 | 5
  Nose: Week 20 | 0 | 0
  Nose: Week 24: number analyzed (Participants) | 5 | 5
  Nose: Week 24 | 0 | 0
  Nose: Week 28: number analyzed (Participants) | 2 | 2
  Nose: Week 28 | 0 | 0
  Nose: Week 32: number analyzed (Participants) | 2 | 3
  Nose: Week 32 | 0 | 0
  Nose: Week 40: number analyzed (Participants) | 1 | 1
  Nose: Week 40 | 0 | 0
  Nose: Week 44: number analyzed (Participants) | 59 | 38
  Nose: Week 44 | 1 | 0
  Skin: Week 18: number analyzed (Participants) | 88 | 84
  Skin: Week 18 | 8 | 4
  Skin: Week 20: number analyzed (Participants) | 4 | 5
  Skin: Week 20 | 3 | 1
  Skin: Week 24: number analyzed (Participants) | 5 | 5
  Skin: Week 24 | 1 | 0
  Skin: Week 28: number analyzed (Participants) | 2 | 2
  Skin: Week 28 | 0 | 0
  Skin: Week 32: number analyzed (Participants) | 2 | 3
  Skin: Week 32 | 0 | 0
  Skin: Week 40: number analyzed (Participants) | 1 | 1
  Skin: Week 40 | 1 | 1
  Skin: Week 44: number analyzed (Participants) | 59 | 38
  Skin: Week 44 | 4 | 2
  Throat: Week 18: number analyzed (Participants) | 88 | 84
  Throat: Week 18 | 4 | 2
  Throat: Week 20: number analyzed (Participants) | 4 | 5
  Throat: Week 20 | 0 | 1
  Throat: Week 24: number analyzed (Participants) | 5 | 5
  Throat: Week 24 | 0 | 0
  Throat: Week 28: number analyzed (Participants) | 2 | 2
  Throat: Week 28 | 0 | 0
  Throat: Week 32: number analyzed (Participants) | 2 | 3
  Throat: Week 32 | 0 | 0
  Throat: Week 40: number analyzed (Participants) | 1 | 1
  Throat: Week 40 | 0 | 0
  Throat: Week 44: number analyzed (Participants) | 59 | 38
  Throat: Week 44 | 0 | 0

69. Secondary Outcome: Open-Label Phase: Number of Participants With Vital Sign Abnormalities
Description: Vital Sign Abnormalities criteria included: sitting diastolic blood pressure millimeters of Mercury (mmHG) of <50 mmHg, sitting pulse rate beats per minute (bpm) of <40 or 120 bpm, sitting systolic blood pressure (mmHG) of <90 mmHg, supine diastolic blood pressure (mmHG) of <50 mmHg, supine pulse rate (BPM) of <40 bpm or >120 bpm, supine systolic blood pressure (mmHG) of 90 mmHg.
Time Frame: From the first dose of study drug up to Week 18
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 225
Participants
  Sitting diastolic BP ([mmHg]): <50 mmHg: number analyzed (Participants) | 219
  Sitting diastolic BP ([mmHg]): <50 mmHg | 0
  Sitting pulse rate (bpm): <40 bpm: number analyzed (Participants) | 219
  Sitting pulse rate (bpm): <40 bpm | 0
  Sitting pulse rate (bpm): >120 bpm: number analyzed (Participants) | 219
  Sitting pulse rate (bpm): >120 bpm | 5
  Sitting systolic BP (mmHg): <90 mmHg: number analyzed (Participants) | 219
  Sitting systolic BP (mmHg): <90 mmHg | 0
  Supine diastolic BP (mmHg): <50 mmHg: number analyzed (Participants) | 28
  Supine diastolic BP (mmHg): <50 mmHg | 2
  Supine pulse rate (bpm): <40 bpm: number analyzed (Participants) | 28
  Supine pulse rate (bpm): <40 bpm | 0
  Supine pulse rate (bpm): >120 bpm: number analyzed (Participants) | 28
  Supine pulse rate (bpm): >120 bpm | 0
  Supine systolic BP (mmHg): <90 mmHg: number analyzed (Participants) | 28
  Supine systolic BP (mmHg): <90 mmHg | 2

70. Secondary Outcome: Double Blind Phase: Number of Participants With Vital Sign Abnormalities
Description: Vital Sign Abnormalities criteria included: diastolic blood pressure (mmHG) of <50 mmHg, Pulse rate (BPM) of <40 bpm or >120 bpm, sitting diastolic blood pressure (mmHG) of <50 mmHg, sitting pulse rate beats per minute (bpm) of <40 bpm or >120 bpm, sitting systolic blood pressure (mmHG) of <90 mmHg, supine diastolic blood pressure (mmHG) of <50 mmHg, supine pulse rate (BPM) of <40 bpm or >120 bpm, supine systolic blood pressure (mmHG) of <90 mmHg, systolic blood pressure (mmHG) of <90 mmHg.
Time Frame: From the first dose of study drug in double blind up to week 44
Population: The DBSAS consists of all participants who have received atleast one dose of study medication in double-blind phase. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure and "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 87 | 82
Participants
  Diastolic BP (mmHg): <50 mmHg: number analyzed (Participants) | 1 | 0
  Diastolic BP (mmHg): <50 mmHg | 0 | 0
  Pulse rate (bpm): <40 bpm: number analyzed (Participants) | 1 | 0
  Pulse rate (bpm): <40 bpm | 0 | 0
  Pulse rate (bpm): >120 bpm: number analyzed (Participants) | 1 | 0
  Pulse rate (bpm): >120 bpm | 0 | 0
  Sitting diastolic BP (mmHg): <50 mmHg: number analyzed (Participants) | 86 | 82
  Sitting diastolic BP (mmHg): <50 mmHg | 0 | 0
  Sitting pulse rate (bpm): <40 bpm: number analyzed (Participants) | 86 | 82
  Sitting pulse rate (bpm): <40 bpm | 0 | 0
  Sitting pulse rate (bpm): >120 bpm: number analyzed (Participants) | 86 | 82
  Sitting pulse rate (bpm): >120 bpm | 0 | 1
  Sitting systolic BP (mmHg): <90 mmHg | 0 | 0
  Supine diastolic BP (mmHg): <50 mmHg: number analyzed (Participants) | 7 | 8
  Supine diastolic BP (mmHg): <50 mmHg | 0 | 0
  Supine pulse rate (bpm): <40 bpm: number analyzed (Participants) | 7 | 8
  Supine pulse rate (bpm): <40 bpm | 0 | 0
  Supine pulse rate (bpm): >120 bpm: number analyzed (Participants) | 7 | 8
  Supine pulse rate (bpm): >120 bpm | 0 | 0
  Supine systolic BP (mmHg): <90 mmHg: number analyzed (Participants) | 7 | 8
  Supine systolic BP (mmHg): <90 mmHg | 1 | 0
  Systolic BP (mmHg): <90 mmHg: number analyzed (Participants) | 1 | 0
  Systolic BP (mmHg): <90 mmHg | 0 | 0

71. Secondary Outcome: Open-Label Phase: Number of Participants With Change From Baseline in Vital Sign Measures
Description: Change in vital Signs included: Sitting diastolic blood pressure [mmHG]: >=20mmHg increase from baseline (IFB) and >= 20mmHg decrease from baseline (DFB). Sitting systolic blood pressure mmHG: >= 30mmHg IFB and >= 30mmHg DFB. Supine diastolic blood pressure mmHG: >= 20mmHg IFB and >= 20mmHg DFB. Supine systolic blood pressure mmHG: >= 30mmHg IFB and >= 30mmHg DFB.
Time Frame: From the first dose of study drug up to Week 18
Population: OLFAS: all participants who were enrolled into OL phase of study and received at least one dose of study medication in open-label phase.Here, 'n' signifies participants evaluable for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Open-Label Phase
Number analyzed (Participants) | 225
Participants
  Sitting diastolic BP: >= 20mmHg IFB: number analyzed (Participants) | 211
  Sitting diastolic BP: >= 20mmHg IFB | 9
  Sitting diastolic BP: >= 20mmHg DFB: number analyzed (Participants) | 211
  Sitting diastolic BP: >= 20mmHg DFB | 14
  Sitting systolic BP: >= 30mmHg IFB: number analyzed (Participants) | 211
  Sitting systolic BP: >= 30mmHg IFB | 2
  Sitting systolic BP: >= 30mmHg DFB: number analyzed (Participants) | 211
  Sitting systolic BP: >= 30mmHg DFB | 5
  Supine diastolic BP: >= 20mmHg IFB: number analyzed (Participants) | 14
  Supine diastolic BP: >= 20mmHg IFB | 0
  Supine diastolic BP: >= 20mmHg DFB: number analyzed (Participants) | 14
  Supine diastolic BP: >= 20mmHg DFB | 3
  Supine systolic BP: >= 30mmHg IFB: number analyzed (Participants) | 14
  Supine systolic BP: >= 30mmHg IFB | 0
  Supine systolic BP: >= 30mmHg DFB: number analyzed (Participants) | 14
  Supine systolic BP: >= 30mmHg DFB | 3

72. Secondary Outcome: Double Blind Phase: Number of Participants With Change From Baseline in Vital Sign Measures
Description: Change in vital Signs included: Sitting diastolic blood pressure (mmHG): >=20mmHg IFB and >= 20mmHg DFB. Sitting systolic blood pressure mmHG: >= 30mmHg IFB and >= 30mmHg DFB. Supine diastolic blood pressure mmHG: >= 20mmHg IFB and >= 20mmHg DFB. Supine systolic blood pressure mmHG: >= 30mmHg IFB and >= 30mmHg DFB.
Time Frame: From the first dose of study drug in double blind up to week 44
Population: The DBSAS consists of all participants who have received at least one dose of study medication in double-blind phase. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure and "n" signifies participants evaluable for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib: Double Blind Phase | Placebo
Number analyzed (Participants) | 87 | 80
Participants
  Sitting diastolic BP: >= 20mmHg IFB: number analyzed (Participants) | 82 | 79
  Sitting diastolic BP: >= 20mmHg IFB | 9 | 3
  Sitting diastolic BP: >= 20mmHg DFB: number analyzed (Participants) | 82 | 79
  Sitting diastolic BP: >= 20mmHg DFB | 7 | 9
  Sitting systolic BP: >= 30mmHg IFB: number analyzed (Participants) | 83 | 79
  Sitting systolic BP: >= 30mmHg IFB | 3 | 4
  Sitting systolic BP: >= 30mmHg DFB: number analyzed (Participants) | 83 | 79
  Sitting systolic BP: >= 30mmHg DFB | 0 | 2
  Supine diastolic BP: >= 20mmHg IFB: number analyzed (Participants) | 4 | 5
  Supine diastolic BP: >= 20mmHg IFB | 0 | 0
  Supine diastolic BP: >= 20mmHg DFB: number analyzed (Participants) | 4 | 5
  Supine diastolic BP: >= 20mmHg DFB | 0 | 0
  Supine systolic BP: >= 30mmHg IFB: number analyzed (Participants) | 4 | 5
  Supine systolic BP: >= 30mmHg IFB | 0 | 0
  Supine systolic BP: >= 30mmHg DFB: number analyzed (Participants) | 4 | 5
  Supine systolic BP: >= 30mmHg DFB | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to week 44
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non serious in another participant or 1 participant may have experienced both serious and non serious event during study.
Arm/Group | Tofacitinib: Open-Label Phase | Tofacitinib: Double Blind Phase | Placebo
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/88 | 0/85
Serious Adverse Events (participants affected / at risk) | 7/225 | 1/88 | 2/85
Other Adverse Events (participants affected / at risk) | 108/225 | 57/88 | 57/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib: Open-Label Phase (N=225) | Tofacitinib: Double Blind Phase (N=88) | Placebo (N=85)
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Condition aggravated (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1
Epidural empyema (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Subperiosteal abscess (Infections and infestations) | 1 | 0 | 0
Still's disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pilonidal sinus repair (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib: Open-Label Phase (N=225) | Tofacitinib: Double Blind Phase (N=88) | Placebo (N=85)
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 1
Uveitis (Eye disorders) | 0 | 0 | 2
Disease progression (General disorders) | 5 | 8 | 13
Pyrexia (General disorders) | 11 | 4 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 8 | 3 | 2
Nasopharyngitis (Infections and infestations) | 10 | 7 | 3
Pharyngitis (Infections and infestations) | 5 | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 5 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 3 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 4 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 24 | 13 | 9
Urinary tract infection (Infections and infestations) | 0 | 1 | 3
Viral infection (Infections and infestations) | 5 | 2 | 1
Alanine aminotransferase increased (Investigations) | 6 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 7 | 4 | 1
Blood creatine phosphokinase increased (Investigations) | 5 | 3 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 2
Haemoglobin decreased (Investigations) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 16 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 2
Vomiting (Gastrointestinal disorders) | 12 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Condition aggravated (General disorders) | 0 | 2 | 2

LIMITATIONS AND CAVEATS:
Data not reported for the PK endpoints, since the PK dataset will be combined together with PK data from other studies and analyze in a pooled analysis; the results of this pooled analysis will be reported separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02592434/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT02592434/SAP_001.pdf